CLINICAL TRIAL: NCT00094302
Title: Treatment of Preserved Cardiac Function Heart Failure With an Aldosterone Antagonist (TOPCAT)
Brief Title: Aldosterone Antagonist Therapy for Adults With Heart Failure and Preserved Systolic Function
Acronym: TOPCAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 160; HHSN268200425207C (Other Grant/Funding Number: NIH contract)
Record Dates: First submitted 2004-10-15; First posted 2004-10-15 (Estimated); Results first posted 2015-03-02 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2014-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Heart Failure, Congestive
Keywords: Heart Failure; Diastolic Heart Failure; Preserved Ejection Fraction
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Heart Failure; Heart Failure, Diastolic | interventions — Spironolactone; Mineralocorticoid Receptor Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo of spironolactone
  Interventions: Drug: Placebo
- Spironolactone (Experimental): Spironolactone (an aldosterone antagonist) is supplied as 15 mg tablets. Drug is taken orally by subjects. The initial study drug dose is 15 mg/day (one tablet) and may be titrated up to 30 mg/day (two tablets) or 45 mg/day (three tablets). Subjects are on study drug for the duration of the trial.
  Interventions: Drug: Spironolactone

INTERVENTIONS:
Drug: Spironolactone — Spironolactone (an aldosterone antagonist) is supplied as 15 mg tablets. Drug is taken orally by subjects. The initial study drug dose is 15 mg/day (one tablet) and may be titrated up to 30 mg/day (two tablets) or 45 mg/day (three tablets). Subjects are on study drug for the duration of the trial.
  Other Names: aldosterone antagonist
  Arms: Spironolactone
Drug: Placebo — Placebo of spironolactone
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness of aldosterone antagonist therapy in reducing cardiovascular mortality, aborted cardiac arrest, and heart failure hospitalization in patients who have heart failure with preserved systolic function.

DETAILED DESCRIPTION:
BACKGROUND:

Heart failure (HF) is a major cause of morbidity and mortality, particularly in older people. Indeed, it is the most common discharge diagnosis in patients older than 65 years. As the United States population ages, heart failure will continue to grow as a public health concern. Therapeutic trials of heart failure have dealt almost exclusively with patients who have systolic dysfunction. However, there is now an emerging awareness that nearly half of the patients with heart failure have preserved systolic function and that the survival of these patients is adversely affected. This study is a randomized clinical trial of a novel therapeutic approach, specifically the use of spironolactone, an aldosterone antagonist, in treating these patients. While this treatment has been shown to be useful in treating heart failure with reduced systolic function, it has not been studied in patients with preserved systolic function.

Patients with heart failure and preserved systolic function have a poor prognosis. The annual mortality rate is intermediate between the prognosis for those without heart failure and for those with heart failure and reduced systolic function. For instance, Family Health Study participants with heart failure and preserved systolic function had a mortality rate of 9% compared to 3% for their age- and gender-matched controls. The mortality rate was 19% in heart failure patients with reduced systolic function heart failure compared to 4% for their matched controls.

As heart failure develops, neurohormones are released that initially improve cardiac output but ultimately contribute to progression of left ventricular dysfunction. The renin-angiotensin-aldosterone system is an important part of this compensatory response. Aldosterone levels may rise to 20 times normal levels in heart failure and aldosterone contributes to the development of myocardial fibrosis. Spironolactone is a potassium-sparing diuretic that acts on the distal tubule, inhibiting sodium and potassium ion exchange. There are several potential beneficial actions, including prevention of cardiac fibrosis. A recent trial evaluated spironolactone in patients with systolic dysfunction heart failure. Spironolactone treatment caused a 30% reduction in mortality compared to placebo (p< 0.001). The improvement resulted from a reduction in all cause mortality. More recently, the Eplerenone Post-Myocardial Infarction (MI) study showed that this aldosterone antagonist significantly reduces mortality despite background treatment with an angiotensin-converting enzyme (ACE) inhibitor and beta-blocker. Advantages of using spironolactone in this study are that it is commercially available, inexpensive, and no longer under patent (therefore this study will not be done by industry). Also, there is a clear physiologic rationale for its use, and the side effect profile is well understood. The study enrolled subjects who had preserved systolic function with heart failure and who met clearly defined eligibility criteria that were selected to make the results widely generalizable to clinical practice.

DESIGN NARRATIVE:

This is a randomized, double-blinded, placebo-controlled trial of aldosterone antagonist therapy (15 mg dose spironolactone or placebo; titrated up to 30 or 45 mg/day) in 3,445 adult patients with heart failure and preserved systolic function. Patients were recruited from August 2006 through January 2012, treated, and will be followed through June 2013. Approximately 270 clinical sites in six countries were subcontracted by the clinical trial coordinating center. Subject visits to a clinical center will occur every four or six months. Data collected include demographic and clinical data, including the results of history and physical exams, laboratory and imaging data, repository specimens for special physiology studies, and genetic studies. Additionally, data regarding quality of life and compliance with assigned treatment will also be collected and assessed.

ELIGIBILITY:
INCLUSION CRITERIA:

* Heart failure as defined by at least one of symptom (paroxysmal nocturnal dyspnea; orthopnea; or dyspnea on mild or moderate exertion) at the time of screening and at least one sign (any rales post cough; jugular venous pressure(JVP) greater than or equal to 10cm of water(H2O); lower extremity edema; or chest x-ray demonstrating pleural effusion, pulmonary congestion, or cardiomegaly) within 12 months prior to study entry:
* left ventricular ejection fraction greater than or equal to 45% (per local reading); the ejection fraction must have been obtained within 6 months prior to randomization and after any MI or other event that would affect ejection fraction
* Controlled systolic blood pressure(BP), defined as a target systolic BP less than 140 mm Hg; participants with BP up to and including 160 mm Hg are eligible for enrollment if they are on three or more medications to control BP
* Serum potassium less than 5.0 mmol/L prior to randomization
* At least one hospital admission for which heart failure was a major component of the hospitalization some time within the 12 months prior to study entry OR brain natriuretic peptide (BNP) greater than or equal to 100pg/ml or N-terminal pro-BNP greater than or equal to 360pg/ml within the 60 days prior to study entry
* Women of child-bearing potential must have a negative serum/urine pregnancy test within 72 hours prior to randomization, must not be lactating, and must agree to use an effective method of contraception during the entire course of study participation
* Willing to comply with scheduled visits
* Informed consent form signed by the subject prior to participation in the trial

EXCLUSION CRITERIA:

* Severe systemic illness with an expected life expectancy of less than 3 years
* Chronic pulmonary disease requiring home O2, oral steroid therapy, or hospitalization for exacerbation within 12 months of study entry, or significant chronic pulmonary disease in the opinion of the investigator
* Known infiltrative or hypertrophic obstructive cardiomyopathy or known pericardial constriction
* Primary hemodynamically significant uncorrected valvular heart disease, obstructive or regurgitant, or any valvular disease expected to lead to surgery during the trial
* Atrial fibrillation with a resting heart rate greater than 90 bpm
* MI in the past 90 days
* Coronary artery bypass graft surgery in the past 90 days
* Percutaneous coronary intervention in the past 30 days
* Heart transplant recipient
* Currently implanted left ventricular assist device
* Stroke in past 90 days
* Systolic BP (SBP) greater than 160 mm Hg
* Known orthostatic hypotension
* Gastrointestinal disorder that could interfere with study drug absorption
* Use of any aldosterone antagonist or potassium sparing medication in the last 14 days or any known condition that would require the use of an aldosterone antagonist during study participation;
* Known intolerance to aldosterone antagonists
* Current lithium use
* Current participation (including prior 30 days) in any other therapeutic trial
* Any condition that, in the opinion of the investigator, may prevent the participant from adhering to the trial protocol
* History of hyperkalemia (serum potassium greater than or equal to 5.5mmol/L) in the past 6 months or serum potassium greater than or equal to 5.0mmol/L within the past 2 weeks
* Severe renal dysfunction, defined as an estimated glomerular filtration rate(GFR) less than 30ml/min. Participants with serum creatinine greater than or equal to 2.5mg/dl are also excluded even if their GFR is greater than or equal to 30ml/min
* Known chronic hepatic disease, defined as aspartate aminotransferase(AST) and alanine aminotransferase(ALT) levels greater than 3.0 times the upper limit of normal as read at the local lab.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3445 (Actual)
Dates: Start 2006-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonja M. McKinlay, PhD, Principal Investigator — New England Research Institutes, Inc.
Locations (270):
- United States (155):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cardiovascular Consultants, Ltd., Glendale, Arizona
  - Carl T. Hayden VA Medical Center, Phoenix, Arizona
  - Central Arkansas Veterans Healthcare System, Little Rock, Arkansas
  - Heart Clinic Arkansas, Little Rock, Arkansas
  - Cynthia Thaik, Burbank, California
  - Fresno VA Medical Center, Fresno, California
  - Clinica Medica San Miguel, Los Angeles, California
  - CAPRI, Los Angeles, California
  - VA Medical Center West Los Angeles, Los Angeles, California
  - Mehrdad Kevin Ariani, MD, Inc., Northridge, California
  - UC Davis Medical Center, Sacremento, California
  - Central Coast Cardiology, Salinas, California
  - Naval Medical Center San Diego, San Diego, California
  - Olive View - UCLA Medial Center, Sylmar, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Cardio-Vascular Institute, Greeley, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Howard University Hospital, Washington D.C., District of Columbia
  - Washington DC VA Hospital, Washington D.C., District of Columbia
  - Daytona Heart Group, Daytona Beach, Florida
  - M & O Clinical Research, LLC, Fort Lauderdale, Florida
  - Florida Heart Center, Ft. Pierce, Florida
  - University of Florida, Gainesville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Brevard Cardiovascular Research Associates, Inc, Rockledge, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Emory University at Grady Health System, Atlanta, Georgia
  - Morehouse School of Medicine, Atlanta, Georgia
  - Northside Cardiology Center, Atlanta, Georgia
  - InnovaMed Alliance, Marietta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois at Chicago Medical Center, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Cardiovascular Research Foundation, Elk Grove Village, Illinois
  - Heart, Lung and Vascular Institute, Peoria, Illinois
  - HeartCare Midwest, Peoria, Illinois
  - The Care Group, LLC, Indianapolis, Indiana
  - Cardiovascular Research of Northwest Indiana, LLC, Munster, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Baptist Healthcare System, Inc. d/b/a Baptist Hospital East, Louisville, Kentucky
  - Leonard J. Chabert Medical Center, Houma, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Northeast Cardiology, Bangor, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Kaiser Permanente, Largo, Maryland
  - Northwest Hospital, Randallstown, Maryland
  - Delmarva Heart Research Foundation, Salisbury, Maryland
  - Associates in Cardiology, PA, Silver Spring, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Caritas St. Elizabeth's Medical Center, Boston, Massachusetts
  - Merrimack Valley Cardiology Associates, Chelmsford, Massachusetts
  - Compass Medical East Bridgewater, East Bridgewater, Massachusetts
  - Pentucket Medical Associates, Haverhill, Massachusetts
  - Charles River Medical Associates, Natick, Massachusetts
  - Hawthorn Medical Associates, North Dartmouth, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Umass Memorial Medical Center, Worcester, Massachusetts
  - Veterans Affairs Ann Arbor Health Care System, Ann Arbor, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Detroit VA Medical Center, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - William Beaumont Health Center, Royal Oak, Michigan
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Heartland Regional Medical Clinic, Saint Joseph, Missouri
  - Glacier View Cardiology, Kalispell, Montana
  - Bryan LGH Heart Institute, Lincoln, Nebraska
  - The Creighton Cardiac Center, Omaha, Nebraska
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Cardiovascular Associates of the Delaware Valley, Elmer, New Jersey
  - Cardiovascular Associates of the Delaware Valley, Haddon Heights, New Jersey
  - NJ Heart, Linden, New Jersey
  - St. Joseph's Regional Medical Center, Paterson, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Electrophysiology Research Foundation, Somerset, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - New Jersey Cardiology Associates, West Orange, New Jersey
  - New York Methodist Hospital, Brooklyn, New York
  - Research Foundation State University of New York at Buffalo, Buffalo, New York
  - Buffalo Heart Group, LLC, Buffalo, New York
  - Jamaica Hospital Medical Center, Jamaica, New York
  - Mid Valley Cardiology, Kingston, New York
  - Winthrop Cardiology Associates, Mineola, New York
  - Soundshore Medical Center of Westchester, New Rochelle, New York
  - NYU School of Medicine, New York, New York
  - St. Lukes Roosevelt, New York, New York
  - Northport VA Medical Center, Northport, New York
  - University of Rochester Medical Center, Rochester, New York
  - Lewin, Fagen, and Lown, MD, PC, Smithtown, New York
  - SUNY Upstate Medical Center, Syracuse, New York
  - Syracuse VA Medical Center, Syracuse, New York
  - Bronx-Lebanon Hospital Center, The Bronx, New York
  - Northeast Medical Center, Concord, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals of Cleveland/Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Hospital East, Columbus, Ohio
  - VAMC Dayton, Dayton, Ohio
  - CCHS Clinical Research Office/Marymount Hospital, Garfield Heights, Ohio
  - CCHS Clinical Research Office/ Hillcrest Hospital, Mayfield Heights, Ohio
  - COR Clinical Research, Oklahoma City, Oklahoma
  - Oklahoma City VA Medical Center, Oklahoma City, Oklahoma
  - Oklahoma Foundation for Cardiovascular Research, Oklahoma City, Oklahoma
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - St. Charles Health System, Bend, Oregon
  - Providence Heart and Vascular Institute, Portland, Oregon
  - Capital Area Research, Camp Hill, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Medicor Associates, Inc, Erie, Pennsylvania
  - The Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster Heart and Stroke Foundation, Lancaster, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital- Dept. of Family and Community Health, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Eastwick Primary Care, Philadelphia, Pennsylvania
  - Pittsburgh VA Healthcare System, Pittsburgh, Pennsylvania
  - The Reading Hospital and Medical Center, West Reading, Pennsylvania
  - Memorial Hospital Rhode Island, Pawtucket, Rhode Island
  - VAMC - Charleston, SC, Charleston, South Carolina
  - Black Hills VA Health Care System, Fort Meade, South Dakota
  - The Stern Cardiovascular Center, Germantown, Tennessee
  - Memphis VA Medical Center, Memphis, Tennessee
  - Memphis Heart Clinic, Memphis, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Vanderbilt Heart and Vascular Institute, Nashville, Tennessee
  - DCT - APHC, LLC dba Discovery Clinical Trials, Arlington, Texas
  - Dallas VA Medical Center, Dallas, Texas
  - Cardiovascular Research Institute of Dallas, Dallas, Texas
  - U.T. Southwestern Medical Center, Dallas, Texas
  - Michael E. DeBakey VA Medical Cntr., Houston, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - Wilford Hall Medical Center, Lackland City, Texas
  - Texas Tech University Health Sciences Center, Odessa, Texas
  - Cardiology Clinic of San Antonio, San Antonio, Texas
  - Tyler Cardiovascular Consultants, Tyler, Texas
  - LDS Hospital, Murray, Utah
  - University of Utah, Salt Lake City, Utah
  - Cardiovascular Associates Ltd., Chesapeake, Virginia
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - Evergreen Healthcare, Kirkland, Washington
  - Providence St. Peter Hospital, Olympia, Washington
  - Sound Health Research, Port Orchard, Washington
  - University of Washington, Seattle, Washington
  - CAMC Health Education and Research Institute, Charleston, West Virginia
  - William S. Middleton Memorial VA Hospital, Madison, Wisconsin
  - University of Wisconsin-Madison, Madison, Wisconsin
  - Aspirus Heart and Vascular Institute, Wausau, Wisconsin
- Argentina (18):
  - Instituto de Investigaciones Clinicas de Bahia Blanca, Bahía Blanca, Buenos Aires
  - IMAI Research, Buenos Aires, Buenos Aires
  - CIPREC, Buenos Aires, Buenos Aires
  - Instituto Cardiologico Ezpecializado S.R.L, Buenos Aires, Buenos Aires
  - Clinica IMA, Buenos Aires, Buenos Aires
  - Clinica Coronel Suarez, Coronel Suárez, Buenos Aires
  - Hospital Italiano de La Plata, La Plata, Buenos Aires
  - Instituto de Investigaciones Clinicas de Mar Del Plata, Mar del Plata, Buenos Aires
  - Instituto de Investigaciones Clinicas de Quilmes, Quilmes, Buenos Aires
  - Clinica Privada Del Prado, Córdoba, Córdoba Province
  - Policlinico Modelo de Cipoletti, Cipolletti, Río Negro Province
  - Hospital San Bernardo, Salta, Salta Province
  - Centro de Investigaciones Clinicas del Litoral SRL, Santa Fe, Santa Fe Province
  - Centro Privado de Cardiologia, San Miguel de Tucumán, Tucumán Province
  - Instituto de Investigaciones Clinicas de Rosario, Rosario Santa Fe
  - Centro Modelo de Cardiología, San Miguel de Tucumán
  - Instituto de Cardiologia SRL, San Miguel de Tucumán
  - Sanatorio Mayo S.A., Santa Fe
- Brazil (17):
  - Hospital Felicio Rocho, Belo Horizonte
  - Santa Casa De Belo Horizonte, Belo Horizonte
  - HMCP PUC Campinas, Campinas
  - Irmandade da Santa Casa de Misericordia de Curitiba, Curitiba Parana
  - Hospital das Clinicas da Universidade Federal de Goias, Goiás
  - Instituto do Coracao de Marilia, Marilia Sao Paulo
  - Hospital Sao Vicente de Paulo, Passo Fundo
  - PROCAPE, Pernambuco
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
  - Hospital Mae De Deus, Porto Alegre
  - Hospital Universitario Pedro Ernesto, Rio de Janeiro
  - Santa Casa de Misericordia do Rio de Janeiro, Rio de Janeiro
  - Instituto de Cardiologia de Santa Catarina, Santa Catarina
  - Incor Fmusp, São Paulo
  - Instituto de Molestias Cardiosvaculares, São Paulo
  - UNIFESP/Hospital Sao Paulo, São Paulo
  - Instituto do Coracao do Triangulo Mineiro, Uberlândia
- Canada (35):
  - University of Calgary, Calgary, Alberta
  - Fraser Clinical Trials Inc., New Westminster, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Health Science Centre, St. John's, Newfoundland and Labrador
  - Capital District Health Authority, Halifax, Nova Scotia
  - Dr. Saul Vizel Cardiac Research Office, Cambridge, Ontario
  - Cornwall Clinical Trials, Cornwall, Ontario
  - Dr. Gurcharan Syan (PP), Greater Sudbury, Ontario
  - Hamilton Health Sciences - General Site, Hamilton, Ontario
  - London Health Sciences Center, London, Ontario
  - Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - CHUS - Hopital Fleurimont, Fleurimont, Quebec
  - Service de la Recherche, Granby, Quebec
  - Cite de la Sante de Laval, Laval, Quebec
  - Clinique Cardiologie Levis, Lévis, Quebec
  - Hopital Du Sacre Coeur de Montreal, Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - CHUM - Hotel Dieu, Montreal, Quebec
  - Chum Hotel Dieu, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Centre de recherche clinique de Quebec, Québec, Quebec
  - C.S.S.S.B., Saint George, Quebec
  - Centre Hosp Regional de Lanaudiere, Sainte Charles Borromee, Quebec
  - Hopital Laval, Ste-Foy, Quebec
  - CSSS du Sud de Lanaudiere (Hopital Pierre-Le Gardeur), Terrebonne, Quebec
  - Centre De Sante et De Services Sociaux De Thetford, Thetford-Mines, Quebec
  - Misericordia Hospital - Cardiac Sciences, Edmonton
  - CDRC Rive-Sud, Longueuil
  - SMBD Jewish General Hospital, Montreal
  - Saskatchewan Heart Centre, Saskatoon
  - Cardiology Clinical Trials - Surrey Memorial Hospital, Surrey
  - Centre Hospitalier de Trois-Rivieres, Trois-Rivières
- Georgia (9):
  - Cardio-Reanimation Centre, Tbilisi, K'alak'i T'bilisi
  - L &J Clinic, Kutaisi
  - Tbilisi State Medical University Clinic #1, Tbilisi
  - Cardiology Clinic, Tbilisi
  - Multiprofile Clinical Hospital of Tbilisi #2, Tbilisi
  - Emergency Cardiology Centre, Tbilisi
  - National Center of Therapy, Tbilisi
  - Diagnostic Services Clinic, Tbilisi
  - Clinic of Angiocardiology "ADAPTI", Tbilisi
- Russia (36):
  - Kaliningrad Region Hospital, Kaliningrad, Kaliningrad Oblast
  - Municipal Healthcare Institution <>, Gatchina, Leningradskaya Oblast'
  - Federal State Institution, Saratov, Saratov Oblast
  - City Healthcare Institution Clinical Hospital #8, Yaroslavl, Yaroslavl Oblast
  - Yaroslavl Regional Clinical Hospital, Yaroslavl, Yaroslavl Oblast
  - Altay State Medical University of federal agency of public health and social progress RF, Barnaul
  - Municipal Health Care Institution "City Hospital #1", Barnaul
  - Kemerovo Cadiologiy Dispensary, Kemerovo Medical Academy, Kemerovo
  - Nonstate Healthcare Institution, Kemerovo
  - State Healthcare Institution "Region Clinical Hospital #1, Krasnodar
  - National Research Center for Preventitive Medicine, Moscow
  - Russian State Medical University, Hospital Therapy Department #1, Moscow
  - State Education High Professional Education Russian State Medical University, Moscow
  - Federal State Institution "Outpatient clinic #3 of President's Management Department of Russian Fede, Moscow
  - Research Institute of Physico-Chemical Medicine Center for Atheosclerosis and Laboratory, Moscow
  - Non State Health Care Institution Central Hospital #6 of Russian Railways JSC, Moscow
  - Novosibirsk Municipal Clinical Emergency Hosp. # 2, Novosibirsk
  - Almasov research institute of Cardiology, Saint Petersberg
  - Public Institution of Health City Hospital # 28, Saint Petersburg
  - State Institution Saint-Petersburg Dzhanelidze Scientific, Saint Petersburg
  - Saint-Petersburg State Healthcare Institution "City Alexander's Hospital", Saint Petersburg
  - Saint-Petersburg Clinical Hospital of RAMS, policlinic department, Saint Petersburg
  - Federal State Health Care Institution, Saint Petersburg
  - Saint-Petersburg State Health Care Institution "City Hospital of Saint George the Martyr", Saint Petersburg
  - Non-state Health Care Institution, Saint Petersburg
  - City Hospital #26, Saint Petersburg
  - City Hospital No 26, Saint Petersburg
  - Chair and Department of Hospital Therapy, Saint Petersburg
  - Medico- Military Academy, Navy Therapy Dept, Saint Petersburg
  - Saint-Petersburg State Institution of Health Protection, "City Hosptial # 15", Saint Petersburg
  - Saint-Petersburg State Health Institution "Pokrovskaya City Hospital", Saint Petersburg
  - Chair of Nephrology and Dialysis of St Petersburg State Medical University, Saint Petersburg
  - State Educational Institution of High Professional Education Saratov State Medical University, Saratov
  - State Institition Research Institution of Cardiology of Tomsk, Tomsk
  - State Educational institution of Higher Professional Education "Volgograd State Medical University o, Volgograd
  - State Health Care Institution "Voronezh Regional Clinical Consultative & Diagnostic Centre", Voronezh

REFERENCES:
- [Background] Desai AS, Lewis EF, Li R, Solomon SD, Assmann SF, Boineau R, Clausell N, Diaz R, Fleg JL, Gordeev I, McKinlay S, O'Meara E, Shaburishvili T, Pitt B, Pfeffer MA. Rationale and design of the treatment of preserved cardiac function heart failure with an aldosterone antagonist trial: a randomized, controlled study of spironolactone in patients with symptomatic heart failure and preserved ejection fraction. Am Heart J. 2011 Dec;162(6):966-972.e10. doi: 10.1016/j.ahj.2011.09.007. Epub 2011 Nov 8. PMID 22137068
- [Result] Shah SJ, Heitner JF, Sweitzer NK, Anand IS, Kim HY, Harty B, Boineau R, Clausell N, Desai AS, Diaz R, Fleg JL, Gordeev I, Lewis EF, Markov V, O'Meara E, Kobulia B, Shaburishvili T, Solomon SD, Pitt B, Pfeffer MA, Li R. Baseline characteristics of patients in the treatment of preserved cardiac function heart failure with an aldosterone antagonist trial. Circ Heart Fail. 2013 Mar;6(2):184-92. doi: 10.1161/CIRCHEARTFAILURE.112.972794. Epub 2012 Dec 20. PMID 23258572
- [Result] Shah AM, Shah SJ, Anand IS, Sweitzer NK, O'Meara E, Heitner JF, Sopko G, Li G, Assmann SF, McKinlay SM, Pitt B, Pfeffer MA, Solomon SD; TOPCAT Investigators. Cardiac structure and function in heart failure with preserved ejection fraction: baseline findings from the echocardiographic study of the Treatment of Preserved Cardiac Function Heart Failure with an Aldosterone Antagonist trial. Circ Heart Fail. 2014 Jan;7(1):104-15. doi: 10.1161/CIRCHEARTFAILURE.113.000887. Epub 2013 Nov 18. PMID 24249049
- [Result] Pitt B, Pfeffer MA, Assmann SF, Boineau R, Anand IS, Claggett B, Clausell N, Desai AS, Diaz R, Fleg JL, Gordeev I, Harty B, Heitner JF, Kenwood CT, Lewis EF, O'Meara E, Probstfield JL, Shaburishvili T, Shah SJ, Solomon SD, Sweitzer NK, Yang S, McKinlay SM; TOPCAT Investigators. Spironolactone for heart failure with preserved ejection fraction. N Engl J Med. 2014 Apr 10;370(15):1383-92. doi: 10.1056/NEJMoa1313731. PMID 24716680
- [Result] Shah AM, Claggett B, Sweitzer NK, Shah SJ, Anand IS, O'Meara E, Desai AS, Heitner JF, Li G, Fang J, Rouleau J, Zile MR, Markov V, Ryabov V, Reis G, Assmann SF, McKinlay SM, Pitt B, Pfeffer MA, Solomon SD. Cardiac structure and function and prognosis in heart failure with preserved ejection fraction: findings from the echocardiographic study of the Treatment of Preserved Cardiac Function Heart Failure with an Aldosterone Antagonist (TOPCAT) Trial. Circ Heart Fail. 2014 Sep;7(5):740-51. doi: 10.1161/CIRCHEARTFAILURE.114.001583. Epub 2014 Aug 13. PMID 25122186
- [Result] Pfeffer MA, Claggett B, Assmann SF, Boineau R, Anand IS, Clausell N, Desai AS, Diaz R, Fleg JL, Gordeev I, Heitner JF, Lewis EF, O'Meara E, Rouleau JL, Probstfield JL, Shaburishvili T, Shah SJ, Solomon SD, Sweitzer NK, McKinlay SM, Pitt B. Regional variation in patients and outcomes in the Treatment of Preserved Cardiac Function Heart Failure With an Aldosterone Antagonist (TOPCAT) trial. Circulation. 2015 Jan 6;131(1):34-42. doi: 10.1161/CIRCULATIONAHA.114.013255. Epub 2014 Nov 18. PMID 25406305
- [Derived] Tang Y, Li W, Wang Z, Chu SH, Wu Y, Jia Z, Hua C, Zhang H, Liu X, Lv Q, Jiang C, Dong JZ, Ma CS, Du X. Changes in frailty based on minimally important difference and the impact of spironolactone on frailty in heart failure with preserved ejection fraction: insights from the TOPCAT trial. Open Heart. 2025 Oct 22;12(2):e003487. doi: 10.1136/openhrt-2025-003487. PMID 41125402
- [Derived] Ferreira JP, Mendonca L, Marques P, Neves JS, Zannad F, Packer M. Albuminuria Is the Key Driver of Kidney Benefit with Aldosterone Receptor Antagonists in Type 2 Diabetes. J Am Soc Nephrol. 2025 Sep 2. doi: 10.1681/ASN.0000000877. Online ahead of print. No abstract available. PMID 40892478
- [Derived] Xu W, Xiao Z, Tang Y, Li Y, Chen X, He F, Huang H, Li C, Liu Y, Zhou J, Wang Y, Bin J, Chen Y. Association of serum potassium time in target range with cardiovascular outcomes in patients with HFpEF. Open Heart. 2025 Aug 21;12(2):e003439. doi: 10.1136/openhrt-2025-003439. PMID 40841122
- [Derived] Xing F, Gao M, Wu Y, Liang W, Jiang J, Dong YG, Li Y, Dong B, Liu C. Influence of depression trajectories in heart failure patients with preserved ejection fractions: a secondary analysis of adverse outcomes in the TOPCAT trial. Heart. 2025 Jul 14;111(15):733-740. doi: 10.1136/heartjnl-2024-324505. PMID 40089312
- [Derived] Fu Y, Feng S, Gu Z, Liu X, Zhu W, Wei B, Guo L. Associations of Depression, Antidepressants with Atrial Fibrillation Risk in HFpEF Patients. Rev Cardiovasc Med. 2024 Oct 22;25(10):370. doi: 10.31083/j.rcm2510370. eCollection 2024 Oct. PMID 39484118
- [Derived] Zhang Q, Tai S, Zhou S. Abdominal obesity is associated with increased worsening renal function risk in patients with heart failure with preserved ejection fraction. BMC Cardiovasc Disord. 2024 Sep 9;24(1):477. doi: 10.1186/s12872-024-04118-0. PMID 39251903
- [Derived] Desai RJ, Glynn RJ, Solomon SD, Claggett B, Wang SV, Vaduganathan M. Individualized Treatment Effect Prediction with Machine Learning - Salient Considerations. NEJM Evid. 2024 Apr;3(4):EVIDoa2300041. doi: 10.1056/EVIDoa2300041. Epub 2024 Mar 26. PMID 38776640
- [Derived] Pfeffer MA, Claggett B. Behind the Scenes of TOPCAT - Bending to Inform. NEJM Evid. 2022 Jan;1(1):EVIDctcs2100007. doi: 10.1056/EVIDctcs2100007. Epub 2022 Jan 10. PMID 38319229
- [Derived] Kondo T, Dewan P, Anand IS, Desai AS, Packer M, Zile MR, Pfeffer MA, Solomon SD, Abraham WT, Shah SJ, Lam CSP, Jhund PS, McMurray JJV. Clinical Characteristics and Outcomes in Patients With Heart Failure: Are There Thresholds and Inflection Points in Left Ventricular Ejection Fraction and Thresholds Justifying a Clinical Classification? Circulation. 2023 Aug 29;148(9):732-749. doi: 10.1161/CIRCULATIONAHA.122.063642. Epub 2023 Jun 27. PMID 37366061
- [Derived] Huang X, Liu X, Jiang Y, Cao Z, Wu M, Chen Z, Sun R, Yu P, Ma J, Zhu W, Chen Y, Wu G, Zhang Y, Wang J. Association of Body Mass Index and Abdominal Obesity with Incidence of Atrial Fibrillation in Heart Failure with Preserved Ejection Fraction. Curr Med Chem. 2025;32(16):3283-3294. doi: 10.2174/0929867330666230606100903. PMID 37282653
- [Derived] Saksena S, Slee A, Natale A, Lakkireddy DR, Shah D, Di Biase L, Lewalter T, Nagarakanti R, Santangeli P. Atrial Fibrillation can adversely impact Heart Failure with Preserved Ejection Fraction by its association with Heart Failure Progression and Mortality: A Post-Hoc Propensity Score-Matched Analysis of the TOPCAT Americas Trial. Europace. 2023 May 19;25(5):euad095. doi: 10.1093/europace/euad095. PMID 37078691
- [Derived] Cao Y, Guo S, Dong Y, Liu C, Zhu W. Comparison of liver fibrosis scores for predicting mortality and morbidity in heart failure with preserved ejection fraction. ESC Heart Fail. 2023 Jun;10(3):1771-1780. doi: 10.1002/ehf2.14336. Epub 2023 Mar 2. PMID 36864701
- [Derived] Curtain JP, Adamson C, Kondo T, Butt JH, Desai AS, Zannad F, Rouleau JL, Rohde LE, Kober L, Anand IS, van Veldhuisen DJ, Zile MR, Lefkowitz MP, Solomon SD, Packer M, Petrie MC, Jhund PS, McMurray JJV. Investigator-reported ventricular arrhythmias and mortality in heart failure with mildly reduced or preserved ejection fraction. Eur Heart J. 2023 Feb 21;44(8):668-677. doi: 10.1093/eurheartj/ehac801. PMID 36632831
- [Derived] Chen C, Zhao J, Xue R, Liu X, Zhu W, Ye M. Prognostic significance of resting cardiac power to left ventricular mass and E/e' ratio in heart failure with preserved ejection fraction. Front Cardiovasc Med. 2022 Aug 18;9:961837. doi: 10.3389/fcvm.2022.961837. eCollection 2022. PMID 36061551
- [Derived] Zhu W, Cao Y, Ye M, Huang H, Wu Y, Ma J, Dong Y, Liu X, Liu C, Lip GYH. Essen Stroke Risk Score Predicts Clinical Outcomes in Heart Failure Patients with Preserved Ejection Fraction: Evidence from the TOPCAT trial. Thromb Haemost. 2023 Jan;123(1):85-96. doi: 10.1055/a-1932-8854. Epub 2022 Aug 29. PMID 36037830
- [Derived] Zeng S, Cai X, Zheng Y, Liu X, Ye M. Associations of body mass index with mortality in heart failure with preserved ejection fraction patients with ischemic versus non-ischemic etiology. Front Cardiovasc Med. 2022 Aug 4;9:966745. doi: 10.3389/fcvm.2022.966745. eCollection 2022. PMID 35990945
- [Derived] Vaduganathan M, Ferreira JP, Rossignol P, Neuen BL, Claggett BL, Pfeffer MA, McMurray JJV, Pitt B, Zannad F, Solomon SD. Effects of steroidal mineralocorticoid receptor antagonists on acute and chronic estimated glomerular filtration rate slopes in patients with chronic heart failure. Eur J Heart Fail. 2022 Sep;24(9):1586-1590. doi: 10.1002/ejhf.2635. Epub 2022 Aug 31. PMID 35867859
- [Derived] Barkoudah E, Claggett BL, Lewis EF, O'Meara E, Clausell N, Diaz R, Fleg JL, Pitt B, Rouleau JL, Solomon SD, Pfeffer MA, Desai AS. Prognostic Impact of Cardiovascular Versus Noncardiovascular Hospitalizations in Heart Failure With Preserved Ejection Fraction: Insights From TOPCAT. J Card Fail. 2022 Sep;28(9):1390-1397. doi: 10.1016/j.cardfail.2022.05.004. Epub 2022 May 28. PMID 35636727
- [Derived] Yang Y, Zhou Y, Cao Y, Dong Y, Liu C, Zhu W. Impact of diabetic retinopathy on prognosis of patients with heart failure with preserved ejection fraction. Nutr Metab Cardiovasc Dis. 2022 Jul;32(7):1711-1718. doi: 10.1016/j.numecd.2022.04.020. Epub 2022 Apr 27. PMID 35606228
- [Derived] Vaduganathan M, Claggett BL, Inciardi RM, Fonarow GC, McMurray JJV, Solomon SD. Estimating the Benefits of Combination Medical Therapy in Heart Failure With Mildly Reduced and Preserved Ejection Fraction. Circulation. 2022 Jun 7;145(23):1741-1743. doi: 10.1161/CIRCULATIONAHA.121.058929. Epub 2022 May 23. No abstract available. PMID 35603667
- [Derived] Ye M, Choy M, Liu X, Huang P, Wu Y, Dong Y, Zhu W, Liu C. Associations of BMI with mortality in HFpEF patients with concomitant diabetes with insulin versus non-insulin treatment. Diabetes Res Clin Pract. 2022 Mar;185:109805. doi: 10.1016/j.diabres.2022.109805. Epub 2022 Feb 24. PMID 35219761
- [Derived] Guo L, Liu X, Yu P, Zhu W. The "Obesity Paradox" in Patients With HFpEF With or Without Comorbid Atrial Fibrillation. Front Cardiovasc Med. 2022 Jan 11;8:743327. doi: 10.3389/fcvm.2021.743327. eCollection 2021. PMID 35087875
- [Derived] Sun J, Tai S, Guo Y, Tang L, Yang H, Li X, Xing Z, Fu L, Zhou S. Sex Differences in Characteristics and Outcomes in Elderly Heart Failure Patients With Preserved Ejection Fraction: A Post-hoc Analysis From TOPCAT. Front Cardiovasc Med. 2021 Oct 4;8:721850. doi: 10.3389/fcvm.2021.721850. eCollection 2021. PMID 34671652
- [Derived] Hejjaji V, Tang Y, Coles T, Jones PG, Reeve BB, Mentz RJ, Spatz ES, Dunlay SM, Caldwell B, Saha A, Tarver ME, Tran A, Patel KK, Henke D, Pina IL, Spertus JA. Psychometric Evaluation of the Kansas City Cardiomyopathy Questionnaire in Men and Women With Heart Failure. Circ Heart Fail. 2021 Sep;14(9):e008284. doi: 10.1161/CIRCHEARTFAILURE.120.008284. Epub 2021 Sep 1. PMID 34465123
- [Derived] Shin SH, Claggett B, Inciardi RM, Santos ABS, Shah SJ, Zile MR, Pfeffer MA, Shah AM, Solomon SD. Prognostic Value of Minimal Left Atrial Volume in Heart Failure With Preserved Ejection Fraction. J Am Heart Assoc. 2021 Aug 3;10(15):e019545. doi: 10.1161/JAHA.120.019545. Epub 2021 Jul 30. PMID 34325519
- [Derived] Li Y, Yu Y, Wu Y, Liang W, Dong B, Xue R, Dong Y, Zhu W, Huang P. Association of Body-Weight Fluctuation With Outcomes in Heart Failure With Preserved Ejection Fraction. Front Cardiovasc Med. 2021 Jun 14;8:689591. doi: 10.3389/fcvm.2021.689591. eCollection 2021. PMID 34195237
- [Derived] Huang P, Guo Z, Liang W, Wu Y, Zhao J, He X, Zhu W, Liu C, Dong Y, Yu Y, Dong B. Weight Change and Mortality Risk in Heart Failure With Preserved Ejection Fraction. Front Cardiovasc Med. 2021 Jun 4;8:681726. doi: 10.3389/fcvm.2021.681726. eCollection 2021. PMID 34150872
- [Derived] Zhu W, Wu Y, Zhou Y, Liang W, Xue R, Wu Z, Wu D, He J, Dong Y, Liu C. Living Alone and Clinical Outcomes in Patients With Heart Failure With Preserved Ejection Fraction. Psychosom Med. 2021 Jun 1;83(5):470-476. doi: 10.1097/PSY.0000000000000945. PMID 33901053
- [Derived] Lin Y, Zhong X, Liu M, Zhang S, Xiong Z, Huang Y, Fan Y, Xu X, Guo Y, Li Y, Sun X, Zhou H, Yang D, Ye X, Liao X, Zhuang X. Risk Stratification and Efficacy of Spironolactone in Patients with Heart Failure with Preserved Ejection Fraction: Secondary Analysis of the TOPCAT Randomized Clinical Trial. Cardiovasc Drugs Ther. 2022 Apr;36(2):323-331. doi: 10.1007/s10557-021-07178-y. Epub 2021 Apr 1. PMID 33791916
- [Derived] De Marco C, Claggett BL, de Denus S, Zile MR, Huynh T, Desai AS, Sirois MG, Solomon SD, Pitt B, Rouleau JL, Pfeffer MA, O'Meara E. Impact of diabetes on serum biomarkers in heart failure with preserved ejection fraction: insights from the TOPCAT trial. ESC Heart Fail. 2021 Apr;8(2):1130-1138. doi: 10.1002/ehf2.13153. Epub 2021 Jan 12. PMID 33438360
- [Derived] Shen L, Jhund PS, Anand IS, Carson PE, Desai AS, Granger CB, Kober L, Komajda M, McKelvie RS, Pfeffer MA, Solomon SD, Swedberg K, Zile MR, McMurray JJV. Developing and validating models to predict sudden death and pump failure death in patients with heart failure and preserved ejection fraction. Clin Res Cardiol. 2021 Aug;110(8):1234-1248. doi: 10.1007/s00392-020-01786-8. Epub 2020 Dec 10. PMID 33301080
- [Derived] Wu Y, Zhu W, He X, Xue R, Liang W, Wei F, Wu Z, Zhou Y, Wu D, He J, Dong Y, Liu C. Influence of polypharmacy on patients with heart failure with preserved ejection fraction: a retrospective analysis on adverse outcomes in the TOPCAT trial. Br J Gen Pract. 2020 Dec 28;71(702):e62-e70. doi: 10.3399/bjgp21X714245. Print 2021 Jan. PMID 33257457
- [Derived] Yang S, Troendle J. Event-specific win ratios and testing with terminal and non-terminal events. Clin Trials. 2021 Apr;18(2):180-187. doi: 10.1177/1740774520972408. Epub 2020 Nov 24. PMID 33231108
- [Derived] Chung EY, Ruospo M, Natale P, Bolignano D, Navaneethan SD, Palmer SC, Strippoli GF. Aldosterone antagonists in addition to renin angiotensin system antagonists for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2020 Oct 27;10(10):CD007004. doi: 10.1002/14651858.CD007004.pub4. PMID 33107592
- [Derived] Zhu W, Liang W, Ye Z, Wu Y, He X, Xue R, Wu Z, Zhou Y, Zhao J, Dong Y, Liu C. Association of physical activity and risk of atrial fibrillation in heart failure with preserved ejection fraction. Nutr Metab Cardiovasc Dis. 2021 Jan 4;31(1):247-253. doi: 10.1016/j.numecd.2020.08.022. Epub 2020 Aug 23. PMID 33097408
- [Derived] Chandra A, Alcala MAD, Claggett B, Desai AS, Fang JC, Heitner JF, Liu J, Pitt B, Solomon SD, Pfeffer MA, Lewis EF. Associations Between Depressive Symptoms and HFpEF-Related Outcomes. JACC Heart Fail. 2020 Dec;8(12):1009-1020. doi: 10.1016/j.jchf.2020.06.010. Epub 2020 Sep 9. PMID 32919912
- [Derived] Zhu W, Wu Y, Zhou Y, Liang W, Xue R, Wu Z, Dong Y, Liu C. CHA2DS2-VASc and ATRIA Scores and Clinical Outcomes in Patients with Heart Failure with Preserved Ejection Fraction. Cardiovasc Drugs Ther. 2020 Dec;34(6):763-772. doi: 10.1007/s10557-020-07011-y. PMID 32583288
- [Derived] Cunningham JW, Vaduganathan M, Claggett BL, John JE, Desai AS, Lewis EF, Zile MR, Carson P, Jhund PS, Kober L, Pitt B, Shah SJ, Swedberg K, Anand IS, Yusuf S, McMurray JJV, Pfeffer MA, Solomon SD. Myocardial Infarction in Heart Failure With Preserved Ejection Fraction: Pooled Analysis of 3 Clinical Trials. JACC Heart Fail. 2020 Aug;8(8):618-626. doi: 10.1016/j.jchf.2020.02.007. Epub 2020 May 6. PMID 32387067
- [Derived] Flint KM, Shah SJ, Lewis EF, Kao DP. Variation in clinical and patient-reported outcomes among complex heart failure with preserved ejection fraction phenotypes. ESC Heart Fail. 2020 Jun;7(3):811-824. doi: 10.1002/ehf2.12660. Epub 2020 Mar 11. PMID 32160420
- [Derived] Myhre PL, Vaduganathan M, O'Meara E, Claggett BL, de Denus S, Jarolim P, Anand IS, Pitt B, Rouleau JL, Solomon SD, Pfeffer MA, Desai AS. Mechanistic Effects of Spironolactone on Cardiovascular and Renal Biomarkers in Heart Failure With Preserved Ejection Fraction: A TOPCAT Biorepository Study. Circ Heart Fail. 2020 Jan;13(1):e006638. doi: 10.1161/CIRCHEARTFAILURE.119.006638. Epub 2020 Jan 20. PMID 31957468
- [Derived] Vardeny O, Claggett B, Vaduganathan M, Beldhuis I, Rouleau J, O'Meara E, Anand IS, Shah SJ, Sweitzer NK, Fang JC, Desai AS, Lewis EF, Pitt B, Pfeffer MA, Solomon SD; TOPCAT Investigators. Influence of Age on Efficacy and Safety of Spironolactone in Heart Failure. JACC Heart Fail. 2019 Dec;7(12):1022-1028. doi: 10.1016/j.jchf.2019.08.019. PMID 31779923
- [Derived] Angraal S, Mortazavi BJ, Gupta A, Khera R, Ahmad T, Desai NR, Jacoby DL, Masoudi FA, Spertus JA, Krumholz HM. Machine Learning Prediction of Mortality and Hospitalization in Heart Failure With Preserved Ejection Fraction. JACC Heart Fail. 2020 Jan;8(1):12-21. doi: 10.1016/j.jchf.2019.06.013. Epub 2019 Oct 9. PMID 31606361
- [Derived] Tromp J, Shen L, Jhund PS, Anand IS, Carson PE, Desai AS, Granger CB, Komajda M, McKelvie RS, Pfeffer MA, Solomon SD, Kober L, Swedberg K, Zile MR, Pitt B, Lam CSP, McMurray JJV. Age-Related Characteristics and Outcomes of Patients With Heart Failure With Preserved Ejection Fraction. J Am Coll Cardiol. 2019 Aug 6;74(5):601-612. doi: 10.1016/j.jacc.2019.05.052. PMID 31370950
- [Derived] Beale AL, Nanayakkara S, Kaye DM. Impact of Sex on Ventricular-Vascular Stiffness and Long-Term Outcomes in Heart Failure With Preserved Ejection Fraction: TOPCAT Trial Substudy. J Am Heart Assoc. 2019 Jul 2;8(13):e012190. doi: 10.1161/JAHA.119.012190. Epub 2019 Jun 22. PMID 31230508
- [Derived] Selvaraj S, Claggett B, Shah SJ, Anand IS, Rouleau JL, Desai AS, Lewis EF, Vaduganathan M, Wang SY, Pitt B, Sweitzer NK, Pfeffer MA, Solomon SD. Utility of the Cardiovascular Physical Examination and Impact of Spironolactone in Heart Failure With Preserved Ejection Fraction. Circ Heart Fail. 2019 Jul;12(7):e006125. doi: 10.1161/CIRCHEARTFAILURE.119.006125. Epub 2019 Jun 21. PMID 31220936
- [Derived] Neefs J, van den Berg NWE, Krul SPJ, Boekholdt SM, de Groot JR. Effect of Spironolactone on Atrial Fibrillation in Patients with Heart Failure with Preserved Ejection Fraction: Post-Hoc Analysis of the Randomized, Placebo-Controlled TOPCAT Trial. Am J Cardiovasc Drugs. 2020 Feb;20(1):73-80. doi: 10.1007/s40256-019-00353-5. PMID 31214914
- [Derived] Kristensen SL, Mogensen UM, Jhund PS, Rorth R, Anand IS, Carson PE, Desai AS, Pitt B, Pfeffer MA, Solomon SD, Zile MR, Kober L, McMurray JJV. N-Terminal Pro-B-Type Natriuretic Peptide Levels for Risk Prediction in Patients With Heart Failure and Preserved Ejection Fraction According to Atrial Fibrillation Status. Circ Heart Fail. 2019 Mar;12(3):e005766. doi: 10.1161/CIRCHEARTFAILURE.118.005766. PMID 30871349
- [Derived] Merrill M, Sweitzer NK, Lindenfeld J, Kao DP. Sex Differences in Outcomes and Responses to Spironolactone in Heart Failure With Preserved Ejection Fraction: A Secondary Analysis of TOPCAT Trial. JACC Heart Fail. 2019 Mar;7(3):228-238. doi: 10.1016/j.jchf.2019.01.003. PMID 30819379
- [Derived] Myhre PL, O'Meara E, Claggett BL, de Denus S, Jarolim P, Anand IS, Beldhuis IE, Fleg JL, Lewis E, Pitt B, Rouleau JL, Solomon SD, Pfeffer MA, Desai AS. Cardiac Troponin I and Risk of Cardiac Events in Patients With Heart Failure and Preserved Ejection Fraction. Circ Heart Fail. 2018 Nov;11(11):e005312. doi: 10.1161/CIRCHEARTFAILURE.118.005312. PMID 30571192
- [Derived] Selvaraj S, Claggett B, Shah SJ, Anand I, Rouleau JL, O'Meara E, Desai AS, Lewis EF, Pitt B, Sweitzer NK, Fang JC, Pfeffer MA, Solomon SD. Prognostic Value of Albuminuria and Influence of Spironolactone in Heart Failure With Preserved Ejection Fraction. Circ Heart Fail. 2018 Nov;11(11):e005288. doi: 10.1161/CIRCHEARTFAILURE.118.005288. PMID 30571191
- [Derived] Myhre PL, Vaduganathan M, Claggett BL, Anand IS, Sweitzer NK, Fang JC, O'Meara E, Shah SJ, Desai AS, Lewis EF, Rouleau J, Pitt B, Pfeffer MA, Solomon SD. Association of Natriuretic Peptides With Cardiovascular Prognosis in Heart Failure With Preserved Ejection Fraction: Secondary Analysis of the TOPCAT Randomized Clinical Trial. JAMA Cardiol. 2018 Oct 1;3(10):1000-1005. doi: 10.1001/jamacardio.2018.2568. PMID 30140899
- [Derived] Cikes M, Claggett B, Shah AM, Desai AS, Lewis EF, Shah SJ, Anand IS, O'Meara E, Rouleau JL, Sweitzer NK, Fang JC, Saksena S, Pitt B, Pfeffer MA, Solomon SD. Atrial Fibrillation in Heart Failure With Preserved Ejection Fraction: The TOPCAT Trial. JACC Heart Fail. 2018 Aug;6(8):689-697. doi: 10.1016/j.jchf.2018.05.005. Epub 2018 Jul 11. PMID 30007557
- [Derived] Lewis EF, Claggett B, Shah AM, Liu J, Shah SJ, Anand I, O'Meara E, Sweitzer NK, Rouleau JL, Fang JC, Desai AS, Retta TM, Solomon SD, Heitner JF, Stamos TD, Boineau R, Pitt B, Pfeffer MA. Racial Differences in Characteristics and Outcomes of Patients With Heart Failure and Preserved Ejection Fraction in the Treatment of Preserved Cardiac Function Heart Failure Trial. Circ Heart Fail. 2018 Mar;11(3):e004457. doi: 10.1161/CIRCHEARTFAILURE.117.004457. PMID 29664406
- [Derived] Vaduganathan M, Claggett BL, Chatterjee NA, Anand IS, Sweitzer NK, Fang JC, O'Meara E, Shah SJ, Hegde SM, Desai AS, Lewis EF, Rouleau J, Pitt B, Pfeffer MA, Solomon SD. Sudden Death in Heart Failure With Preserved Ejection Fraction: A Competing Risks Analysis From the TOPCAT Trial. JACC Heart Fail. 2018 Aug;6(8):653-661. doi: 10.1016/j.jchf.2018.02.014. Epub 2018 Mar 4. PMID 29501806
- [Derived] Rossignol P, Claggett BL, Liu J, Vardeny O, Pitt B, Zannad F, Solomon S. Spironolactone and Resistant Hypertension in Heart Failure With Preserved Ejection Fraction. Am J Hypertens. 2018 Mar 10;31(4):407-414. doi: 10.1093/ajh/hpx210. PMID 29228101
- [Derived] Selvaraj S, Claggett B, Shah SJ, Anand I, Rouleau JL, Desai AS, Lewis EF, Pitt B, Sweitzer NK, Pfeffer MA, Solomon SD. Systolic blood pressure and cardiovascular outcomes in heart failure with preserved ejection fraction: an analysis of the TOPCAT trial. Eur J Heart Fail. 2018 Mar;20(3):483-490. doi: 10.1002/ejhf.1060. Epub 2017 Nov 16. PMID 29148144
- [Derived] Pokharel Y, Khariton Y, Tang Y, Nassif ME, Chan PS, Arnold SV, Jones PG, Spertus JA. Association of Serial Kansas City Cardiomyopathy Questionnaire Assessments With Death and Hospitalization in Patients With Heart Failure With Preserved and Reduced Ejection Fraction: A Secondary Analysis of 2 Randomized Clinical Trials. JAMA Cardiol. 2017 Dec 1;2(12):1315-1321. doi: 10.1001/jamacardio.2017.3983. PMID 29094152
- [Derived] Hegde SM, Claggett B, Shah AM, Lewis EF, Anand I, Shah SJ, Sweitzer NK, Fang JC, Pitt B, Pfeffer MA, Solomon SD. Physical Activity and Prognosis in the TOPCAT Trial (Treatment of Preserved Cardiac Function Heart Failure With an Aldosterone Antagonist). Circulation. 2017 Sep 12;136(11):982-992. doi: 10.1161/CIRCULATIONAHA.117.028002. Epub 2017 Jun 21. PMID 28637881
- [Derived] Anand IS, Claggett B, Liu J, Shah AM, Rector TS, Shah SJ, Desai AS, O'Meara E, Fleg JL, Pfeffer MA, Pitt B, Solomon SD. Interaction Between Spironolactone and Natriuretic Peptides in Patients With Heart Failure and Preserved Ejection Fraction: From the TOPCAT Trial. JACC Heart Fail. 2017 Apr;5(4):241-252. doi: 10.1016/j.jchf.2016.11.015. PMID 28359411
- [Derived] Biering-Sorensen T, Shah SJ, Anand I, Sweitzer N, Claggett B, Liu L, Pitt B, Pfeffer MA, Solomon SD, Shah AM. Prognostic importance of left ventricular mechanical dyssynchrony in heart failure with preserved ejection fraction. Eur J Heart Fail. 2017 Aug;19(8):1043-1052. doi: 10.1002/ejhf.789. Epub 2017 Mar 21. PMID 28322009
- [Derived] Santos AB, Roca GQ, Claggett B, Sweitzer NK, Shah SJ, Anand IS, Fang JC, Zile MR, Pitt B, Solomon SD, Shah AM. Prognostic Relevance of Left Atrial Dysfunction in Heart Failure With Preserved Ejection Fraction. Circ Heart Fail. 2016 Apr;9(4):e002763. doi: 10.1161/CIRCHEARTFAILURE.115.002763. PMID 27056882
- [Derived] Joseph J, Claggett BC, Anand IS, Fleg JL, Huynh T, Desai AS, Solomon SD, O'Meara E, Mckinlay S, Pitt B, Pfeffer MA, Lewis EF. QRS Duration Is a Predictor of Adverse Outcomes in Heart Failure With Preserved Ejection Fraction. JACC Heart Fail. 2016 Jun;4(6):477-86. doi: 10.1016/j.jchf.2016.02.013. Epub 2016 Mar 30. PMID 27039126
- [Derived] Lewis EF, Kim HY, Claggett B, Spertus J, Heitner JF, Assmann SF, Kenwood CT, Solomon SD, Desai AS, Fang JC, McKinlay SA, Pitt BA, Pfeffer MA; TOPCAT Investigators. Impact of Spironolactone on Longitudinal Changes in Health-Related Quality of Life in the Treatment of Preserved Cardiac Function Heart Failure With an Aldosterone Antagonist Trial. Circ Heart Fail. 2016 Mar;9(3):e001937. doi: 10.1161/CIRCHEARTFAILURE.114.001937. PMID 26962133
- [Derived] Shah AM, Claggett B, Sweitzer NK, Shah SJ, Deswal A, Anand IS, Fleg JL, Pitt B, Pfeffer MA, Solomon SD. Prognostic Importance of Changes in Cardiac Structure and Function in Heart Failure With Preserved Ejection Fraction and the Impact of Spironolactone. Circ Heart Fail. 2015 Nov;8(6):1052-8. doi: 10.1161/CIRCHEARTFAILURE.115.002249. Epub 2015 Oct 16. PMID 26475142
- [Derived] Solomon SD, Claggett B, Lewis EF, Desai A, Anand I, Sweitzer NK, O'Meara E, Shah SJ, McKinlay S, Fleg JL, Sopko G, Pitt B, Pfeffer MA; TOPCAT Investigators. Influence of ejection fraction on outcomes and efficacy of spironolactone in patients with heart failure with preserved ejection fraction. Eur Heart J. 2016 Feb 1;37(5):455-62. doi: 10.1093/eurheartj/ehv464. Epub 2015 Sep 15. PMID 26374849
- [Derived] Shah AM, Claggett B, Sweitzer NK, Shah SJ, Anand IS, Liu L, Pitt B, Pfeffer MA, Solomon SD. Prognostic Importance of Impaired Systolic Function in Heart Failure With Preserved Ejection Fraction and the Impact of Spironolactone. Circulation. 2015 Aug 4;132(5):402-14. doi: 10.1161/CIRCULATIONAHA.115.015884. Epub 2015 Jun 30. PMID 26130119
- [Derived] Borlaug BA, Lewis GD, McNulty SE, Semigran MJ, LeWinter M, Chen H, Lin G, Deswal A, Margulies KB, Redfield MM. Effects of sildenafil on ventricular and vascular function in heart failure with preserved ejection fraction. Circ Heart Fail. 2015 May;8(3):533-41. doi: 10.1161/CIRCHEARTFAILURE.114.001915. Epub 2015 Mar 17. PMID 25782985
- [Derived] Hamo CE, Heitner JF, Pfeffer MA, Kim HY, Kenwood CT, Assmann SF, Solomon SD, Boineau R, Fleg JL, Spertus JA, Lewis EF. Baseline distribution of participants with depression and impaired quality of life in the Treatment of Preserved Cardiac Function Heart Failure with an Aldosterone Antagonist Trial. Circ Heart Fail. 2015 Mar;8(2):268-77. doi: 10.1161/CIRCHEARTFAILURE.114.001838. Epub 2015 Feb 3. PMID 25648577
- [Derived] Mak GJ, Ledwidge MT, Watson CJ, Phelan DM, Dawkins IR, Murphy NF, Patle AK, Baugh JA, McDonald KM. Natural history of markers of collagen turnover in patients with early diastolic dysfunction and impact of eplerenone. J Am Coll Cardiol. 2009 Oct 27;54(18):1674-82. doi: 10.1016/j.jacc.2009.08.021. PMID 19850207
- See also: Link to PubMed ID #25406305 publication in Circulation — http://circ.ahajournals.org/content/early/2014/11/18/CIRCULATIONAHA.114.013255.long

RESULTS

PARTICIPANT FLOW:
Recruitment Details: TOPCAT enrolled 3445 patients with heart failure and preserved ejection fraction at 233 academic and community medical centers in 6 countries between August 2006 and January 2012. Trial follow-up ended in June 2013.
Pre-assignment Details: Trial randomization was stratified by whether patients were enrolled into the study on the basis of having a hospitalization for heart failure within the past year (N=2,464) or having an elevated natriuretic peptide level within 60 days before randomization (N=981). The second criterion was considered only for those who did not meet the first.
Period: Overall Study
Arm/Group | Placebo | Spironolactone
Started | 1723 | 1722
Completed | 1306 | 1316
Not Completed | 417 | 406
Not completed — Lost to Follow-up | 43 | 41
Not completed — Physician Decision | 5 | 8
Not completed — Withdrawal by Subject | 103 | 111
Not completed — Death | 266 | 246

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Spironolactone | Total
Number analyzed (Participants) | 1723 | 1722 | 3445
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 649 | 654 | 1303
  >=65 years | 1074 | 1068 | 2142
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68.7 [60.7 to 75.5] | 68.7 [61.0 to 76.4] | 68.7 [60.9 to 75.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 887 | 888 | 1775
  Male | 836 | 834 | 1670
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 6 | 9
  Asian | 9 | 10 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 149 | 151 | 300
  White | 1537 | 1525 | 3062
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 25 | 28 | 53
Region of Enrollment [Number; unit: participants]
  United States | 579 | 572 | 1151
  Canada | 160 | 166 | 326
  Argentina | 60 | 63 | 123
  Brazil | 82 | 85 | 167
  Russian Federation | 537 | 529 | 1066
  Georgia | 305 | 307 | 612
Eligibility Stratum [Number; unit: participants] — Eligible patients were assigned to one of two strata before randomization, according to whether they had at least one hospitalization within the previous 12 months in which management of heart failure was a major component of the care provided, or in absence of that criterion, an elevated brain natriuretic peptide (BNP) level within 60 days prior to randomization (a brain natriuretic peptide [BNP] level ≥100 pg per milliliter or an N-terminal pro-BNP [NTproBNP] level ≥360 pg per milliliter).
  participants
    Hospitalization in previous year for heart failure | 1232 | 1232 | 2464
    Elevated natriuretic peptide in previous 60 days | 491 | 490 | 981

OUTCOME MEASURES:

1. Primary Outcome: Composite Outcome of Cardiovascular Mortality, Aborted Cardiac Arrest, or Hospitalization for the Management of Heart Failure, Whichever Occurred First
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 6 years per subject.
Population: All Participants who were randomized were included in the analysis. The analysis was Intention to Treat, meaning all participants were analyzed based on their initial treatment assignment and not on the treatment eventually received.
Measure: Number; unit: Events per 100 person-years
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 1723 | 1722
Events per 100 person-years | 6.6 | 5.9
Statistical Analysis 1: Comparison: Placebo vs Spironolactone; Composite endpoint was compared by trial arm using logrank test of time to first event from time of randomization. Time to event was the time at which the first observed event component of the composite endpoint was observed. This endpoint was adjudicated by the TOPCAT clinical endpoints committee. There were 320 subjects in the Spironolactone group and 351 subjects in Placebo group with a confirmed event. Subjects who did not experience this endpoint were censored at time of last contact; Test type: Superiority or Other; p = 0.14, Log Rank — No covariate adjustment; Two-sided log rand test (0.05 Type 1 error); Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.77 to 1.04] — Spironolactone compared to Placebo

2. Secondary Outcome: Cardiovascular Mortality
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 6 years per subject.
Population: as for outcome 1
Measure: Number; unit: Events per 100 person-years
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 1723 | 1722
Events per 100 person-years | 3.1 | 2.8
Statistical Analysis 1: Comparison: Placebo vs Spironolactone; This endpoint was compared by trial arm (spironolactone vs. placebo) using a logrank test of time to event from the time of randomization. Subjects who did not experience this endpoint were censored at the time of their last contact. This endpoint was adjudicated by the TOPCAT clinical endpoints committee. There were 336 subjects (160 in the Spironolactone group and 176 in the Placebo group) with a confirmed event; Test type: Superiority or Other; p = 0.35, Log Rank — No covariate adjustment; Two-sided log rand test (0.05 Type 1 error); Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.73 to 1.12] — Spironolactone compared to Placebo

3. Secondary Outcome: Aborted Cardiac Arrest
Description: First incidence of aborted cardiac arrest
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 6 years per subject.
Population: as for outcome 1
Measure: Number; unit: Events per 100 person-years
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 1723 | 1722
Events per 100 person-years | 0.09 | 0.05
Statistical Analysis 1: Comparison: Placebo vs Spironolactone; This endpoint was compared by trial arm (spironolactone vs. placebo) using a logrank test of time to first event from the time of randomization. Subjects who did not experience this endpoint were censored at the time of their last contact. This endpoint was adjudicated by the TOPCAT clinical endpoints committee. There were 8 subjects (3 in the Spironolactone group and 5 in the Placebo group) with a confirmed event; Test type: Superiority or Other; p = 0.48, Log Rank — No covariate adjustment; Two-sided log rand test (0.05 Type 1 error); Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.14 to 2.50] — Spironolactone compared to Placebo

4. Secondary Outcome: Hospitalization for the Management of Heart Failure
Description: First incidence of a hospitalization for the management of heart failure
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 6 years per subject.
Population: as for outcome 1
Measure: Number; unit: Events per 100 person-years
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 1723 | 1722
Events per 100 person-years | 4.6 | 3.8
Statistical Analysis 1: Comparison: Placebo vs Spironolactone; This endpoint was compared by trial arm (spironolactone vs. placebo) using a logrank test of time to first event from the time of randomization. Subjects who did not experience this endpoint were censored at the time of their last contact. This endpoint was adjudicated by the TOPCAT clinical endpoints committee. There were 451 subjects (206 in the Spironolactone group and 245 in the Placebo group) who have been confirmed to have experienced the event; Test type: Superiority or Other; p = 0.04, Log Rank — No covariate adjustment; Two-sided log rand test (0.05 Type 1 error); Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.69 to 0.99] — Spironolactone compared to Placebo

5. Secondary Outcome: All-cause Mortality
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 6 years per subject.
Population: as for outcome 1
Measure: Number; unit: Events per 100 person-years
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 1723 | 1722
Events per 100 person-years | 4.6 | 4.2
Statistical Analysis 1: Comparison: Placebo vs Spironolactone; Endpoint compared by trial arm using logrank test of time to event from randomization. Subjects who did not experience endpoint were censored at time of last contact. Attempts were made to determine vital status as of each subject's last potential visit, based on randomization, even if the subject ended study participation before then. This outcome was adjudicated. There were 252 events over 6,022 patient-years in Spironolactone arm and 274 events over 5,981 patient-years in Placebo arm; Test type: Superiority or Other; p = 0.29, Log Rank — No covariate adjustment; Two-sided log rand test (0.05 Type 1 error); Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.77 to 1.08] — Spironolactone compared to Placebo

6. Secondary Outcome: Composite Outcome of Cardiovascular Mortality or Cardiovascular-related Hospitalization (i.e., Hospitalization for Myocardial Infarction(MI), Stroke, or the Management of Heart Failure), Whichever Occurred First
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 6 years per subject.
Population: as for outcome 1
Measure: Number; unit: Events per 100 person-years
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 1723 | 1722
Events per 100 person-years | 7.8 | 7.2
Statistical Analysis 1: Comparison: Placebo vs Spironolactone; Composite endpoint was compared by trial arm using logrank test of time to first event from time of randomization. Time to event was the time at which the first observed event component of the composite endpoint was observed. Component endpoints were adjudicated by the TOPCAT clinical endpoints committee. There were 382 subjects in Spironolactone group and 404 subjects in Placebo group with a confirmed event. Subjects who did not experience this endpoint were censored at time of last contact; Test type: Superiority or Other; p = 0.28, Log Rank — No covariate adjustment; Two-sided log rank test (0.05 Type 1 error); Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.80 to 1.06] — Spironolactone compared to Placebo

7. Secondary Outcome: Cardiovascular-related Hospitalization
Description: Hospitalization for MI, stroke or the management of heart failure, whichever occurred first
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 6 years per subject.
Population: as for outcome 1
Measure: Number; unit: Events per 100 person-years
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 1723 | 1722
Events per 100 person-years | 6.2 | 5.5
Statistical Analysis 1: Comparison: Placebo vs Spironolactone; Endpoint was compared by trial arm using logrank test of time to first event from time of randomization. Time to event was the time at which the first observed event component of the composite endpoint was observed. Component endpoints were adjudicated by the TOPCAT clinical endpoints committee. There were 291 subjects in Spironolactone group and 320 subjects in Placebo group with a confirmed event. Subjects who did not experience this endpoint were censored at time of last contact; Test type: Superiority or Other; p = 0.15, Log Rank — No covariate adjustment; Two-sided log rank test (0.05 Type 1 error); Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.76 to 1.04] — Spironolactone compared to Placebo

8. Secondary Outcome: Total Hospitalizations (Including Repeat Hospitalizations) for the Management of Heart Failure
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 6 years per subject.
Population: as for outcome 1
Measure: Number; unit: Events per 100 person-years
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 1723 | 1722
Events per 100 person-years | 8.3 | 6.8
Statistical Analysis 1: Comparison: Placebo vs Spironolactone; There were a total of 869 confirmed heart failure hospitalizations (394 in the Spironolactone group and 475 in the Placebo group) during the 11,471 person-years collected over the course of the TOPCAT trial (5,755 person-years in the Spironolactone group and 5,716 person-years in the Placebo group). The incidence rate of heart failure hospitalizations for each treatment group was compared using a negative binomial regression with a p-value threshold of 0.05 for statistical significance; Test type: Superiority or Other; p = 0.03, Negative binomial regression — No covariate adjustment; incidence rate ratio = 0.75, 95% CI 2-sided [0.58 to 0.97] — Spironolactone compared to Placebo

9. Secondary Outcome: Composite Outcome of Sudden Death or Aborted Cardiac Arrest, Whichever Occurred First
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 6 years per subject.
Population: as for outcome 1
Measure: Number; unit: Events per 100 person-years
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 1723 | 1722
Events per 100 person-years | 1.1 | 1.0
Statistical Analysis 1: Comparison: Placebo vs Spironolactone; Composite endpoint was compared by trial arm using logrank test of time to first event from time of randomization. Time to event was the time at which the first observed event component of the composite endpoint was observed. Component endpoints were adjudicated by the TOPCAT clinical endpoints committee. There were 58 subjects in the Spironolactone group and 60 subjects in Placebo group with a confirmed event. Subjects who did not experience this endpoint were censored at time of last contact; Test type: Superiority or Other; p = 0.82, Log Rank — No covariate adjustment; Two-sided log rank test (0.05 Type 1 error); Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.67 to 1.38] — Spironolactone compared to Placebo

10. Secondary Outcome: New Onset Diabetes Mellitus, Among Subjects Without a History of Diabetes Mellitus at Baseline.
Description: First incidence of new onset diabetes mellitus among subjects without a history of diabetes mellitus at baseline.
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 6 years per subject.
Population: All Participants who were randomized and did not have a history of diabetes mellitus at baseline were included in the analysis. The analysis was Intention to Treat, meaning all participants were analyzed based on their initial treatment assignment and not on the treatment eventually received.
Measure: Number; unit: Events per 100 person-years
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 1167 | 1156
Events per 100 person-years | 0.7 | 0.7
Statistical Analysis 1: Comparison: Placebo vs Spironolactone; This endpoint was compared by trial arm (spironolactone vs. placebo) using a logrank test of time to first event from the time of randomization. Subjects who did not experience this endpoint were censored at the time of their last contact. This endpoint was adjudicated by the TOPCAT clinical endpoints committee. There were 56 subjects (29 in the Spironolactone group and 27 in the Placebo group) with confirmed events; Test type: Superiority or Other; p = 0.76, Log Rank — No covariate adjustment; Two-sided log rank test (0.05 Type 1 error); Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.64 to 1.83] — Spironolactone compared to Placebo

11. Secondary Outcome: Development of Atrial Fibrillation, Among Subjects Without a History of Atrial Fibrillation at Baseline.
Description: First incidence of atrial fibrillation among subjects without a history of atrial fibrillation at baseline
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 6 years per subject.
Population: All Participants who were randomized and did not have a history of atrial fibrillation at baseline were included in the analysis. The analysis was Intention to Treat, meaning all participants were analyzed based on their initial treatment assignment and not on the treatment eventually received.
Measure: Number; unit: Events per 100 person-years
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 1117 | 1111
Events per 100 person-years | 1.4 | 1.4
Statistical Analysis 1: Comparison: Placebo vs Spironolactone; This endpoint was compared by trial arm (spironolactone vs. placebo) using a logrank test of time to first event from the time of randomization. Subjects who did not experience this endpoint were censored at the time of their last contact. This endpoint was adjudicated by the TOPCAT clinical endpoints committee. There were 103 subjects (52 in the Spironolactone group and 51 in the Placebo group) with confirmed events; Test type: Superiority or Other; p = 0.94, Log Rank — No covariate adjustment; Two-sided log rank test (0.05 Type 1 error); Hazard Ratio, log = 1.02, 95% CI 2-sided [0.69 to 1.50] — Spironolactone compared to Placebo

12. Secondary Outcome: Myocardial Infarction
Description: First incidence of myocardial infarction
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 6 years per subject.
Population: as for outcome 1
Measure: Number; unit: Events per 100 person-years
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 1723 | 1722
Events per 100 person-years | 1.1 | 1.2
Statistical Analysis 1: Comparison: Placebo vs Spironolactone; This endpoint was compared by trial arm (spironolactone vs. placebo) using a logrank test of time to first event from the time of randomization. Subjects who did not experience this endpoint were censored at the time of their last contact. This endpoint was adjudicated by the TOPCAT clinical endpoints committee. There were 129 subjects (65 in the Spironolactone group and 64 in the Placebo group) with confirmed events; Test type: Superiority or Other; p = 0.98, Log Rank — No covariate adjustment; Two-sided log rand test (0.05 Type 1 error); Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.71 to 1.42] — Spironolactone compared to Placebo

13. Secondary Outcome: Stroke
Description: First incidence of stroke
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 6 years per subject.
Population: as for outcome 1
Measure: Number; unit: Events per 100 person-years
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 1723 | 1722
Events per 100 person-years | 1.1 | 1.0
Statistical Analysis 1: Comparison: Placebo vs Spironolactone; This endpoint was compared by trial arm (spironolactone vs. placebo) using a logrank test of time to first event from the time of randomization. Subjects who did not experience this endpoint were censored at the time of their last contact. This endpoint was adjudicated by the TOPCAT clinical endpoints committee. There were 117 subjects (57 in the Spironolactone group and 60 in the Placebo group) with confirmed events; Test type: Superiority or Other; p = 0.73, Log Rank — No covariate adjustment; Two-sided log rand test (0.05 Type 1 error); Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.65 to 1.35] — Spironolactone compared to Placebo

14. Secondary Outcome: Deterioration of Renal Function
Description: First incidence of a deterioration of renal function. The TOPCAT protocol defines deterioration of renal function as occurring if a subject has a serum creatinine value which is at least double the baseline value for that subject, and is also above the upper limit of normal (assumed to be 1.0 mg/dL for females and 1.2 mg/dL for males.)
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 6 years per subject.
Population: as for outcome 1
Measure: Number; unit: Events per 100 person-years
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 1723 | 1722
Events per 100 person-years | 2.2 | 3.2
Statistical Analysis 1: Comparison: Placebo vs Spironolactone; This endpoint was compared by trial arm (spironolactone vs. placebo) using a logrank test of time to first event from the time of randomization. Subjects who did not experience this endpoint were censored at the time of their last contact. There were 295 subjects (175 in the Spironolactone group and 120 in the Placebo group) experiencing this endpoint. This endpoint did not undergo adjudication by the TOPCAT clinical endpoints committee; Test type: Superiority or Other; p < 0.01, Log Rank — No covariate adjustment; Two-sided log rand test (0.05 Type 1 error); Hazard Ratio (HR) = 1.49, 95% CI 2-sided [1.18 to 1.87] — Spironolactone compared to Placebo

15. Secondary Outcome: Composite Outcome of Sudden Death, Aborted Cardiac Arrest, or Hospitalization for the Management of Ventricular Tachycardia, Whichever Occurred First
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 6 years per subject.
Population: as for outcome 1
Measure: Number; unit: Events per 100 person-years
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 1723 | 1722
Events per 100 person-years | 1.1 | 1.0
Statistical Analysis 1: Comparison: Placebo vs Spironolactone; Composite endpoint was compared by trial arm using logrank test of time to first event from time of randomization. Time to event was the time at which the first observed event component of the composite endpoint was observed. Component endpoints were adjudicated by the TOPCAT clinical endpoints committee. There were 58 subjects in the Spironolactone group and 61 subjects in Placebo group with a confirmed event. Subjects who did not experience this endpoint were censored at time of last contact; Test type: Superiority or Other; p = 0.75, Log Rank — No covariate adjustment; Two-sided log rank test (0.05 Type 1 error); Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.66 to 1.35] — Spironolactone compared to Placebo

16. Secondary Outcome: Quality of Life, as Measured by the Kansas City Cardiomyopathy Questionnaire.
Description: Average post-baseline quality of life, taking into consideration baseline quality of life, treatment group, the time between the post-baseline measures, and the correlation between repeated measures within an individual.
  The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. Scores are transformed to a range of 0-100, in which higher scores reflect better health status. The KCCQ was administered at the following study visits: baseline, month 4, month 12 and annually thereafter.
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 6 years per subject.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 1723 | 1722
units on a scale | 63.1 (0.3) | 64.4 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Spironolactone; A generalized linear model was fit, with the post-baseline quality of life scores as the dependent variable, and the baseline quality of life score, treatment group, month of visit, and the interaction between treatment group and month of visit as predictor variables. This tests whether the slope of the post-baseline quality of life parameter differs by treatment group, taking into account that measurements in the same subject over time may be correlated; Test type: Superiority or Other; p = 0.27, Regression, Linear
Statistical Analysis 2: Comparison: Placebo vs Spironolactone; Since the p-value for the preceding test (Statistical Analysis 1) was not significant at the 0.05 level, another generalized linear model was fit, omitting the interaction between treatment group and month of visit. This tests whether the value of the post-baseline quality of life parameter differs by treatment group, taking into account that measurements in the same subject over time may be correlated; Test type: Superiority or Other; p < 0.01, Regression, Linear

17. Secondary Outcome: Quality of Life, as Measured by the EuroQOL Visual Analog Scale.
Description: Average post-baseline quality of life, taking into consideration baseline quality of life, treatment group, the time between the post-baseline measures, and the correlation between repeated measures within an individual.
  The EuroQOL visual analog scale (EQ5D) is a single-item, self-administered instrument that quantifies current health status. Scores can range from 0-100, in which higher scores reflect better health status. The EQ5D was administered at the following study visits: baseline, month 4, month 12 and annually thereafter.
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 6 years per subject.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 1723 | 1722
units on a scale | 65.9 (0.3) | 66.4 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Spironolactone; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.87, Regression, Linear
Statistical Analysis 2: Comparison: Placebo vs Spironolactone; [analysis description as in outcome 16, analysis 2]; Test type: Superiority or Other; p = 0.16, Regression, Linear

18. Secondary Outcome: Quality of Life, as Measured by McMaster Overall Treatment Evaluation Questionnaire.
Description: Average post-baseline quality of life, taking into consideration baseline quality of life and treatment group.
  The McMaster Overall Treatment Evaluation questionnaire is a self-administered 3-item instrument that measures a patient's perception of change in their health-related quality of life since the start of therapy. The questionnaire consists of a single question - "Since treatment started, has there been any change in your activity limitation, symptoms and/or feelings related to your heart condition?" Scores can range from -7 to +7, and higher scores reflect better health status. The questionnaire was administered at the following study visits: month 4 and month 12. Valid translations of this questionnaire were only available for subjects enrolled in the United States, Canada and Argentina.
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 6 years per subject.
Population: All Participants from United States, Canada and Argentina who were randomized were included in the analysis. The analysis was Intention to Treat, meaning all participants were analyzed based on their initial treatment assignment and not on the treatment eventually received.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 799 | 801
units on a scale | 1.2 (0.1) | 1.2 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Spironolactone; A generalized linear model was fit, with the post-baseline quality of life scores as the dependent variable, and the baseline quality of life score and treatment group as predictor variables. This tests whether the value of the post-baseline quality of life parameter differs by treatment group; Test type: Superiority or Other; p = 0.99, Regression, Linear

19. Secondary Outcome: Depression Symptoms, as Measured by Patient Health Questionnaire.
Description: Average post-baseline depression, taking into consideration baseline depression, treatment group, the time between the post-baseline measures, and the correlation between repeated measures within an individual.
  The Patient Health Questionnaire (PHQ) is a 10-item, self-administered instrument for screening, diagnosing, monitoring and measuring the severity of depression. Scores can range from 0-27, in which lower scores reflect better mental health status. The PH-Q was administered at the following study visits: baseline, month 12 and annually thereafter. Valid translations of this questionnaire were only available for subjects enrolled in the United States and Canada.
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 6 years per subject.
Population: All Participants from the United States and Canada who were randomized were included in the analysis. The analysis was Intention to Treat, meaning all participants were analyzed based on their initial treatment assignment and not on the treatment eventually received.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 739 | 738
units on a scale | 5.6 (0.1) | 5.1 (0.2)
Statistical Analysis 1: Comparison: Placebo vs Spironolactone; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.39, Regression, Linear
Statistical Analysis 2: Comparison: Placebo vs Spironolactone; [analysis description as in outcome 16, analysis 2]; Test type: Superiority or Other; p = 0.01, Regression, Linear

20. Secondary Outcome: Hospitalization for Any Reason
Description: First incidence of a hospitalization for any reason
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 6 years per subject.
Population: as for outcome 1
Measure: Number; unit: Events per 100 person-years
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 1723 | 1722
Events per 100 person-years | 20.0 | 18.8
Statistical Analysis 1: Comparison: Placebo vs Spironolactone; This endpoint was compared by trial arm (spironolactone vs. placebo) using a logrank test of time to first event from the time of randomization. Subjects who did not experience this endpoint were censored at the time of their last contact. There were a total of 1558 subjects (766 subjects in the Spironolactone group and 792 subjects in the Placebo) who were hospitalized for any cause while on study. This endpoint was not adjudicated by the TOPCAT clinical endpoints committee; Test type: Superiority or Other; p = 0.25, Log Rank — No covariate adjustment; Two-sided log rand test (0.05 Type 1 error); Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.85 to 1.04] — Spironolactone compared to Placebo

21. Secondary Outcome: Potassium
Description: Average post-baseline Potassium, taking into consideration baseline Potassium, treatment group, the time between the post-baseline measures, and the correlation between repeated measures within an individual.
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 6 years per subject.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mEq/L
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 1723 | 1722
mEq/L | 4.32 (0.01) | 4.49 (0.01)
Statistical Analysis 1: Comparison: Placebo vs Spironolactone; A generalized linear model was fit, with the post-baseline laboratory value as the dependent variable, and the baseline laboratory value, treatment group, month of visit, and the interaction between treatment group and month of visit as predictor variables. This tests whether the slope of the post-baseline laboratory parameter differs by treatment group, taking into account that measurements in the same subject over time may be correlated; Test type: Superiority or Other; p = 0.27, Regression, Linear
Statistical Analysis 2: Comparison: Placebo vs Spironolactone; Since the p-value for the preceding test (Statistical Analysis 1) was not significant at the 0.05 level, another generalized linear model was fit, omitting the interaction between treatment group and month of visit. This tests whether the value of the post-baseline laboratory parameter differs by treatment group, taking into account that measurements in the same subject over time may be correlated; Test type: Superiority or Other; p < 0.01, Regression, Linear

22. Secondary Outcome: Serum Creatinine
Description: Average post-baseline serum creatinine, taking into consideration baseline serum creatinine, treatment group, the time between the post-baseline measures, and the correlation between repeated measures within an individual.
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 6 years per subject.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 1723 | 1722
mg/dL | 1.11 (0.005) | 1.17 (0.01)
Statistical Analysis 1: Comparison: Placebo vs Spironolactone; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; p = 0.53, Regression, Linear
Statistical Analysis 2: Comparison: Placebo vs Spironolactone; [analysis description as in outcome 21, analysis 2]; Test type: Superiority or Other; p < 0.01, Regression, Linear

23. Secondary Outcome: Sodium
Description: Average post-baseline Sodium, taking into consideration baseline Sodium, treatment group, the time between the post-baseline measures, and the correlation between repeated measures within an individual.
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 6 years per subject.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mEq/L
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 1723 | 1722
mEq/L | 140.95 (0.06) | 140.33 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Spironolactone; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; p = 0.11, Regression, Linear
Statistical Analysis 2: Comparison: Placebo vs Spironolactone; [analysis description as in outcome 21, analysis 2]; Test type: Superiority or Other; p < 0.01, Regression, Linear

24. Secondary Outcome: Chloride
Description: Average post-baseline Chloride, taking into consideration baseline Chloride, treatment group, the time between the post-baseline measures, and the correlation between repeated measures within an individual.
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 6 years per subject.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mEq/L
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 1723 | 1722
mEq/L | 102.33 (0.08) | 102.26 (0.08)
Statistical Analysis 1: Comparison: Placebo vs Spironolactone; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; p = 0.59, Regression, Linear
Statistical Analysis 2: Comparison: Placebo vs Spironolactone; [analysis description as in outcome 21, analysis 2]; Test type: Superiority or Other; p = 0.54, Regression, Linear

25. Secondary Outcome: Estimated Glomerular Filtration Rate (GFR)
Description: Average post-baseline GFR, taking into consideration baseline GFR, treatment group, the time between the post-baseline measures, and the correlation between repeated measures within an individual.
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 6 years per subject.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73m2
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 1723 | 1722
mL/min/1.73m2 | 67.50 (0.29) | 65.20 (0.90)
Statistical Analysis 1: Comparison: Placebo vs Spironolactone; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; p = 0.98, Regression, Linear
Statistical Analysis 2: Comparison: Placebo vs Spironolactone; [analysis description as in outcome 21, analysis 2]; Test type: Superiority or Other; p = 0.02, Regression, Linear

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) include any untoward medical occurrence which occurred after a subject gave informed consent and no later than 30 days after a subject permanently discontinued the study medication, for a maximum of 6 years per subject.
Description: If a subject experiences more than 1 of a given AE within a system organ class (SOC), the subject was counted only once for that AE.
Arm/Group | Placebo | Spironolactone
Serious Adverse Events (participants affected / at risk) | 855/1723 | 835/1722
Other Adverse Events (participants affected / at risk) | 1086/1723 | 1152/1722
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=1723) | Spironolactone (N=1722)
ABDOMINAL AORTIC ANEURYSM (Cardiac disorders) | 1 (1) | 0 (0)
ABDOMINAL AORTIC ANEURYSM (Vascular disorders) | 2 (2) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 7 (7) | 10 (10)
ABDOMINAL PAIN (Hepatobiliary disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ABDOMINAL VISCUS PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABNORMAL ELECTROLYTE (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ABNORMAL LAB VALUE (Cardiac disorders) | 0 (0) | 1 (1)
ABNORMAL VAGINAL BLEEDING (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ABNORMAL VAGINAL BLEEDING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ABSCESS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ABSCESS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ABSCESS (Surgical and medical procedures) | 0 (0) | 1 (1)
ACID REFLUX (Gastrointestinal disorders) | 0 (0) | 1 (1)
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 9 (9) | 11 (11)
ACUTE MENIERE'S DISEASE (Ear and labyrinth disorders) | 1 (1) | 0 (0)
ACUTE RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
ADRENAL INSUFFIENCY (Endocrine disorders) | 1 (1) | 0 (0)
ALCOHOL WITHDRAWAL (General disorders) | 0 (0) | 1 (1)
ALLERGY (Immune system disorders) | 1 (1) | 0 (0)
ALTERED MENTAL STATUS (Nervous system disorders) | 9 (9) | 8 (8)
ALVEOLITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ALZHEIMER'S DISEASE (Nervous system disorders) | 0 (0) | 2 (2)
AMYLOIDOSIS (Cardiac disorders) | 0 (0) | 1 (1)
AMYLOIDOSIS (Immune system disorders) | 1 (1) | 0 (0)
AMYOTROPHIC LATERAL SCLEROSIS (Nervous system disorders) | 1 (1) | 0 (0)
ANAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ANEMIA (Blood and lymphatic system disorders) | 23 (26) | 15 (18)
ANEMIA (Gastrointestinal disorders) | 2 (3) | 2 (2)
ANEURYSM (Cardiac disorders) | 0 (0) | 1 (1)
ANEURYSM (Vascular disorders) | 3 (3) | 0 (0)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
ANGIOGRAPHY (Cardiac disorders) | 0 (0) | 1 (1)
ANGIOPLASTY (Cardiac disorders) | 0 (0) | 2 (2)
ANXIETY (Nervous system disorders) | 2 (2) | 0 (0)
AORTIC ANEURYSM (Cardiac disorders) | 1 (1) | 1 (1)
AORTIC ANEURYSM (Vascular disorders) | 0 (0) | 1 (1)
AORTIC REGURGITATION (Cardiac disorders) | 0 (0) | 1 (1)
AORTIC STENOSIS (Cardiac disorders) | 2 (2) | 5 (5)
APPENDECTOMY (Surgical and medical procedures) | 0 (0) | 2 (2)
APPENDICEAL ABCESS (Gastrointestinal disorders) | 1 (1) | 0 (0)
APPENDICITIS (Gastrointestinal disorders) | 5 (5) | 1 (1)
ARM INJURY (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
ARM INJURY (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
ARM INJURY (Vascular disorders) | 1 (1) | 0 (0)
ARRHYTHMIA (Cardiac disorders) | 6 (6) | 6 (6)
ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 (0) | 2 (2)
ARTERIAL STENOSIS (Cardiac disorders) | 1 (2) | 2 (2)
ARTERIAL STENOSIS (Renal and urinary disorders) | 0 (0) | 1 (1)
ARTERIAL THROMBOSIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
ARTERIAL THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
ARTHROPLASTY (Surgical and medical procedures) | 0 (0) | 1 (1)
ASCITES (Gastrointestinal disorders) | 0 (0) | 1 (1)
ASCITES (General disorders) | 0 (0) | 1 (1)
ASCITES (Hepatobiliary disorders) | 0 (0) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 5 (6)
ATAXIA (Nervous system disorders) | 2 (2) | 0 (0)
ATHEROSCLEROSIS (Cardiac disorders) | 3 (3) | 1 (1)
ATHEROSCLEROSIS (Vascular disorders) | 2 (2) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 58 (69) | 73 (92)
ATRIAL FIBRILLATION (Renal and urinary disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ATRIAL FLUTTER (Cardiac disorders) | 6 (10) | 8 (10)
AV BLOCK (Cardiac disorders) | 2 (2) | 3 (3)
AV REPLACEMENT (Cardiac disorders) | 1 (1) | 1 (1)
AV STENOSIS (Cardiac disorders) | 1 (1) | 1 (1)
AZOTEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
BACK INJURY (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
BACK PAIN (Cardiac disorders) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 10 (12)
BACTERIAL INFECTION (Infections and infestations) | 0 (0) | 2 (2)
BARIATRIC SURGERY (Gastrointestinal disorders) | 1 (1) | 0 (0)
BELLS PALSY (Nervous system disorders) | 1 (1) | 0 (0)
BI BLEED (Gastrointestinal disorders) | 0 (0) | 1 (1)
BILE DUCT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BILIARY COLIC (Hepatobiliary disorders) | 1 (1) | 0 (0)
BINODAL DISEASE (Cardiac disorders) | 0 (0) | 1 (1)
BIPOLAR DISORDER (Psychiatric disorders) | 0 (0) | 1 (1)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BLADDER OBSTRUCTION (Renal and urinary disorders) | 2 (2) | 0 (0)
BLEEDING IN EYE (Eye disorders) | 0 (0) | 1 (3)
BLISTERS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BLOOD IN STOOL (Gastrointestinal disorders) | 0 (0) | 2 (2)
BLURRED VISION (Eye disorders) | 1 (1) | 0 (0)
BODY PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BOWEL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 5 (6)
BOWEL OBSTRUCTION (Gastrointestinal disorders) | 5 (7) | 7 (7)
BOWEL PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 10 (11) | 9 (9)
BRAIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BRAIN CANCER (Nervous system disorders) | 1 (1) | 1 (1)
BRAIN HEMORRHAGE (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
BRAIN HEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
BRAIN HEMORRHAGE (Nervous system disorders) | 3 (4) | 1 (1)
BRAIN TUMOR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 3 (4)
BREAST REDUCTION (Surgical and medical procedures) | 1 (1) | 0 (0)
BREAST TUMOR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BRONCHIECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 11 (12)
BRUISE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BUTTOCK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
C-DIFF INFECTION (Infections and infestations) | 3 (3) | 2 (2)
CABG (Cardiac disorders) | 0 (0) | 2 (2)
CABG (Surgical and medical procedures) | 0 (0) | 2 (2)
CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 12 (12) | 10 (10)
CARDIAC ARRYTHMIA (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC CATHETERIZATION (Cardiac disorders) | 1 (1) | 1 (1)
CARDIAC CIRRHOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
CARDIAC TAMPONADE (Cardiac disorders) | 1 (1) | 0 (0)
CARDIO RENAL SYNDROME (Cardiac disorders) | 1 (1) | 0 (0)
CARDIOGENIC SHOCK (Cardiac disorders) | 4 (5) | 3 (3)
CARDIOMYOPATHY (Cardiac disorders) | 3 (4) | 2 (2)
CARDIOPULMONARY ARREST (Cardiac disorders) | 2 (2) | 5 (5)
CARDIOSCLEROSIS (Cardiac disorders) | 1 (1) | 1 (1)
CAROTID STENOSIS (Cardiac disorders) | 1 (1) | 1 (1)
CAROTID STENOSIS (Vascular disorders) | 1 (1) | 0 (0)
CAROTID STENT (Surgical and medical procedures) | 1 (1) | 0 (0)
CATARACTS (Eye disorders) | 5 (7) | 5 (7)
CELLULITIS (Infections and infestations) | 14 (14) | 13 (14)
CELLULITIS (Skin and subcutaneous tissue disorders) | 21 (25) | 14 (17)
CENTRAL CHORIORETINAL DYSTROPHY (Eye disorders) | 1 (1) | 1 (1)
CHEST PAIN (Cardiac disorders) | 144 (186) | 143 (203)
CHEST PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
CHEST PAIN (Investigations) | 1 (1) | 0 (0)
CHEST PAIN (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (8)
CHEST PAIN (Renal and urinary disorders) | 0 (0) | 1 (1)
CHOLANGIOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
CHOLANGITIS (Hepatobiliary disorders) | 1 (1) | 1 (1)
CHOLE (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLECYSTECTOMY (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLECYSTECTOMY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CHOLECYSTECTOMY (Surgical and medical procedures) | 0 (0) | 2 (2)
CHOLECYSTITIS (Hepatobiliary disorders) | 10 (11) | 7 (7)
CHOLECYSTITIS (Renal and urinary disorders) | 2 (2) | 0 (0)
CHOLESTASIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHOLESTATIC SYNDROME (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHOPPED WOUND OF LEFT HAND (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CHORIORRETINOPATHY (Eye disorders) | 0 (0) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Cardiac disorders) | 1 (1) | 1 (3)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Renal and urinary disorders) | 1 (1) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 21 (24) | 23 (32)
CIRRHOSIS (Hepatobiliary disorders) | 1 (2) | 1 (1)
COLD EXTREMITIES (Vascular disorders) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 6 (6) | 3 (3)
COLON CANCER (Gastrointestinal disorders) | 0 (0) | 2 (2)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 3 (3)
CONFUSION (Nervous system disorders) | 4 (4) | 1 (1)
CONGESTIVE HEART FAILURE (Cardiac disorders) | 0 (0) | 2 (3)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 2 (2)
CORONAROGRAPHY (Surgical and medical procedures) | 0 (0) | 1 (1)
CORONARY ANGIOGRAPHY (Surgical and medical procedures) | 0 (0) | 1 (1)
CORONARY ARTERY BYPASS GRAFT (Cardiac disorders) | 2 (2) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 17 (18) | 15 (15)
CORONARY ARTERY STENT (Cardiac disorders) | 0 (0) | 1 (1)
CORONARY REVASCULARIZATION (Cardiac disorders) | 0 (0) | 1 (1)
CORONARY VASOSPASM (Cardiac disorders) | 0 (0) | 1 (1)
CORRECTION THERAPY (Surgical and medical procedures) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
COUMADIN TOXICITY (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
CROHNS DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0)
DEATH (Cardiac disorders) | 3 (3) | 4 (4)
DEATH (General disorders) | 83 (84) | 71 (71)
DEATH (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
DEATH (Nervous system disorders) | 0 (0) | 1 (1)
DECREASED APPETITE (Gastrointestinal disorders) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 6 (7) | 4 (5)
DEHYDRATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
DEHYDRATION (General disorders) | 8 (8) | 7 (7)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
DEMENTIA (Nervous system disorders) | 1 (1) | 0 (0)
DENATURED ALCOHOL POISONING (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
DENTAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 3 (5)
DESTABILIZATION OF BLOOD PRESSURE (Cardiac disorders) | 0 (0) | 1 (1)
DEVICE CHANGE (Cardiac disorders) | 6 (6) | 5 (5)
DEVICE IMPLANT (Cardiac disorders) | 1 (1) | 0 (0)
DEVICE MALFUNCTION (Cardiac disorders) | 3 (3) | 0 (0)
DIABETES (Endocrine disorders) | 6 (6) | 14 (17)
DIARRHEA (Cardiac disorders) | 1 (1) | 0 (0)
DIARRHEA (Gastrointestinal disorders) | 7 (8) | 5 (6)
DILATED ESOPHAGUS (Gastrointestinal disorders) | 0 (0) | 1 (1)
DISCITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
DIVERTICULITIS (Gastrointestinal disorders) | 3 (3) | 2 (2)
DIVERTICULOSIS (Gastrointestinal disorders) | 0 (0) | 2 (3)
DIZZINESS (General disorders) | 3 (3) | 5 (5)
DIZZINESS (Nervous system disorders) | 0 (0) | 3 (3)
DORSOPATHY (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
DRUG OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
DRUG TOXOCITY (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
DRY EYES (Eye disorders) | 1 (1) | 0 (0)
DYSARTHRIA (Nervous system disorders) | 1 (1) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 3 (3) | 0 (0)
DYSPHAGIA (Nervous system disorders) | 0 (0) | 1 (1)
DYSPNEA (Cardiac disorders) | 11 (12) | 11 (13)
DYSPNEA (Renal and urinary disorders) | 0 (0) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
EDEMA (Cardiac disorders) | 1 (1) | 0 (0)
EDEMA (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
ELECTIVE BAND PROCEDURE (Gastrointestinal disorders) | 1 (1) | 0 (0)
ELECTROLYTE IMBALANCE (General disorders) | 0 (0) | 1 (1)
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ELEVATED CARDIAC ENZYMES (Cardiac disorders) | 3 (3) | 2 (2)
ELEVATED CREATININE (Renal and urinary disorders) | 1 (1) | 5 (5)
ELEVATED INR (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
ELEVATED LIVER ENZYMES (Hepatobiliary disorders) | 1 (1) | 0 (0)
ELEVATED PT (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
EMBOLECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
ENCEPHALITIS (Infections and infestations) | 0 (0) | 1 (1)
ENCEPHALOPATHY (Hepatobiliary disorders) | 3 (3) | 1 (3)
ENCEPHALOPATHY (Nervous system disorders) | 5 (6) | 8 (8)
ENDARTERECTOMY (Surgical and medical procedures) | 1 (1) | 1 (1)
ENDOCARDITIS (Cardiac disorders) | 0 (0) | 3 (3)
ENDOSCOPIC RETROGRADE CHOLANGIO-PANCREATOGRAPHY (Gastrointestinal disorders) | 1 (1) | 0 (0)
ENTERITIS (Cardiac disorders) | 1 (1) | 0 (0)
ENTEROCOLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
EPIDIDYMITIS (Reproductive system and breast disorders) | 0 (0) | 3 (4)
EPIGASTRIC PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
EPISTAXIS (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
EPISTAXIS (Vascular disorders) | 1 (1) | 2 (3)
EQUIPMENT MALFUNCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 (0) | 1 (1)
EROSION OF PACEMAKER POCKET (Cardiac disorders) | 0 (0) | 1 (1)
EROSION OF THE VAGINAL EPITHELIUM (Reproductive system and breast disorders) | 1 (1) | 0 (0)
ESOPHAGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
ESOPHAGITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
EXACERBATION OF THE CHRONIC CALCULOUS CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
EXTRASYSTOLE (Cardiac disorders) | 2 (2) | 0 (0)
EYE LESION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
EYE SURGERY (Eye disorders) | 1 (1) | 1 (2)
FAILURE TO THRIVE (Cardiac disorders) | 0 (0) | 1 (1)
FAILURE TO THRIVE (General disorders) | 6 (6) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FALL (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (7)
FALL (Nervous system disorders) | 1 (1) | 1 (1)
FASCIOTOMY (Surgical and medical procedures) | 1 (2) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 2 (2)
FECAL IMPACTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
FEMORAL EMBOLUS (Vascular disorders) | 1 (1) | 0 (0)
FEVER (General disorders) | 1 (1) | 2 (2)
FISTULA (Gastrointestinal disorders) | 0 (0) | 1 (1)
FISTULA (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
FOOT INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FOOT PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
FOOT ULCER (Vascular disorders) | 1 (1) | 0 (0)
FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
FRACTURE (Musculoskeletal and connective tissue disorders) | 39 (41) | 31 (34)
GALLSTONES (Hepatobiliary disorders) | 10 (11) | 6 (6)
GANGRENE (Infections and infestations) | 2 (2) | 1 (1)
GANGRENE (Vascular disorders) | 1 (1) | 4 (4)
GASTRECTOMY (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRIC BYPASS SURGERY (Gastrointestinal disorders) | 1 (1) | 2 (2)
GASTRIC BYPASS SURGERY (Surgical and medical procedures) | 0 (0) | 1 (1)
GASTRIC REFLUX (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 3 (3)
GASTROENTERITIS (Gastrointestinal disorders) | 3 (3) | 7 (7)
GASTROPARESIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GATRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GENERAL HEALTH DECLINE (General disorders) | 0 (0) | 3 (3)
GERD (Gastrointestinal disorders) | 0 (0) | 1 (1)
GI BLEED (Gastrointestinal disorders) | 22 (30) | 25 (26)
GI DISTRESS (Gastrointestinal disorders) | 2 (2) | 1 (1)
GOUT (Musculoskeletal and connective tissue disorders) | 6 (11) | 6 (6)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
GUILLIAN BARRE SYNDROME (Immune system disorders) | 1 (2) | 0 (0)
GYNECOMASTIA (Endocrine disorders) | 0 (0) | 1 (1)
GYNECOMASTIA (Reproductive system and breast disorders) | 0 (0) | 1 (2)
HAND PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
HEAD INJURY (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
HEAD INJURY (Nervous system disorders) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1) | 5 (5)
HEARING LOSS (Nervous system disorders) | 0 (0) | 1 (1)
HEART (Cardiac disorders) | 0 (0) | 1 (1)
HEART BLOCK (Cardiac disorders) | 1 (1) | 0 (0)
HEART FAILURE (Cardiac disorders) | 294 (532) | 256 (465)
HEART FAILURE (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
HEART FAILURE (Endocrine disorders) | 0 (0) | 1 (1)
HEART FAILURE (Infections and infestations) | 0 (0) | 1 (1)
HEART FAILURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
HEART FAILURE (Renal and urinary disorders) | 1 (1) | 1 (1)
HEART FAILURE (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
HEART SURGERY (Surgical and medical procedures) | 1 (1) | 0 (0)
HEARTBURN (Cardiac disorders) | 2 (2) | 0 (0)
HEAT (Cardiac disorders) | 0 (0) | 1 (1)
HEEL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
HEMATOCHEZIA (Gastrointestinal disorders) | 2 (2) | 0 (0)
HEMATOMA (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
HEMATOMA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
HEMATOMA (Nervous system disorders) | 3 (3) | 1 (1)
HEMATOMA (Vascular disorders) | 0 (0) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 4 (4) | 5 (5)
HEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
HEMORRHAGE (Gastrointestinal disorders) | 2 (2) | 3 (3)
HEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0)
HEMORRHAGE (Vascular disorders) | 0 (0) | 1 (1)
HEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 0 (0)
HEPARIN BRIDGING (Surgical and medical procedures) | 1 (1) | 0 (0)
HEPATIC ENCEPHALOPATHY (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATOMEGALY (Hepatobiliary disorders) | 0 (0) | 1 (1)
HERNIA (Cardiac disorders) | 1 (1) | 0 (0)
HERNIA (Gastrointestinal disorders) | 3 (3) | 1 (1)
HERNIA (Infections and infestations) | 1 (1) | 0 (0)
HERNIA (Musculoskeletal and connective tissue disorders) | 3 (3) | 8 (10)
HERNIA (Surgical and medical procedures) | 1 (1) | 0 (0)
HERNIATED DISC (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
HIATAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
HIP PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
HIP REPLACEMENT (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
HIP REPLACEMENT (Surgical and medical procedures) | 1 (1) | 0 (0)
HOSPITALIZATION (Cardiac disorders) | 0 (0) | 2 (2)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 1 (1)
HYPERCALCEMIA (General disorders) | 0 (0) | 2 (2)
HYPERCAPNIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPEREMIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
HYPERGLYCEMIA (Endocrine disorders) | 2 (4) | 9 (10)
HYPERKALEMIA (Cardiac disorders) | 0 (0) | 1 (1)
HYPERKALEMIA (Renal and urinary disorders) | 5 (5) | 20 (21)
HYPERNATREMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
HYPERTENSION (Cardiac disorders) | 21 (24) | 27 (32)
HYPERTENSION (General disorders) | 0 (0) | 1 (1)
HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPERTHYROIDISM (Endocrine disorders) | 1 (1) | 1 (1)
HYPERVOLEMIA (Cardiac disorders) | 3 (3) | 1 (1)
HYPERVOLEMIA (General disorders) | 1 (1) | 1 (1)
HYPOGLYCEMIA (Endocrine disorders) | 4 (4) | 7 (8)
HYPOKALEMIA (Renal and urinary disorders) | 4 (5) | 0 (0)
HYPONATREMIA (Endocrine disorders) | 0 (0) | 1 (1)
HYPONATREMIA (General disorders) | 0 (0) | 1 (1)
HYPONATREMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
HYPONATREMIA (Renal and urinary disorders) | 1 (1) | 2 (2)
HYPOTENSION (Cardiac disorders) | 18 (18) | 17 (18)
HYPOTENSION (Endocrine disorders) | 1 (1) | 0 (0)
HYPOVENTILATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPOVOLEMIA (Cardiac disorders) | 1 (1) | 0 (0)
HYPOVOLEMIA (Renal and urinary disorders) | 0 (0) | 2 (2)
HYPOXEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
HYSTERECTOMY (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ICD IMPLANTATION (Surgical and medical procedures) | 1 (1) | 0 (0)
ICD MALFUNCTION (Cardiac disorders) | 1 (1) | 2 (2)
ILEITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
ILEUS (Gastrointestinal disorders) | 1 (1) | 1 (1)
IN-STENT RESTENOSIS (Cardiac disorders) | 1 (2) | 0 (0)
INCREASE THIGH MASS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
INCREASING NITRONGENATED SCORIAS (Renal and urinary disorders) | 0 (0) | 1 (1)
INFECTION (Infections and infestations) | 3 (3) | 3 (4)
INFECTION (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
INFLUENZA (Infections and infestations) | 1 (1) | 1 (1)
INTESTINAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTRACRANIAL BLEED (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
JAUNDICE (Hepatobiliary disorders) | 1 (1) | 0 (0)
KIDNEY DISEASE (Cardiac disorders) | 5 (6) | 4 (4)
KIDNEY DISEASE (General disorders) | 0 (0) | 1 (1)
KIDNEY DISEASE (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
KIDNEY DISEASE (Renal and urinary disorders) | 51 (68) | 63 (79)
KIDNEY DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
KIDNEY FAILURE (Renal and urinary disorders) | 0 (0) | 1 (1)
KIDNEY INFECTION (Renal and urinary disorders) | 1 (1) | 0 (0)
KIDNEY STONE (Renal and urinary disorders) | 2 (2) | 3 (3)
KNEE AMPUTATION (Vascular disorders) | 0 (0) | 1 (1)
KNEE ARTHROPLASTY (Surgical and medical procedures) | 0 (0) | 1 (1)
KNEE INJURY (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
KNEE PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
KNEE SURGERY (Surgical and medical procedures) | 4 (4) | 3 (3)
LABYRINTHITIS (Ear and labyrinth disorders) | 1 (1) | 0 (0)
LARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LARYNGEAL EDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
LEG AMPUTATION (Surgical and medical procedures) | 0 (0) | 1 (1)
LEG CLAUDICATION (Vascular disorders) | 1 (1) | 0 (0)
LEG INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LEG PAIN (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
LEG ULCERS (Vascular disorders) | 1 (1) | 0 (0)
LESION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
LEUKEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
LEUKEMIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
LEUKEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
LIMB ISCHEMIA (Vascular disorders) | 1 (1) | 1 (1)
LIVER CANCER (Hepatobiliary disorders) | 1 (1) | 0 (0)
LIVER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (2)
LIVER LACERATION (Hepatobiliary disorders) | 0 (0) | 1 (1)
LOWER EXTREMITY EDEMA (Cardiac disorders) | 1 (1) | 1 (1)
LOWER EXTREMITY ISCHEMIA (Cardiac disorders) | 0 (0) | 1 (1)
LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 9 (9)
LUNG CONTUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
LYMPHANGITIS (Vascular disorders) | 1 (1) | 0 (0)
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (11) | 0 (0)
MALLORY-WEISS SYNDROME (Gastrointestinal disorders) | 0 (0) | 1 (1)
MALNUTRITION (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
MEDICAL EXAM (Cardiac disorders) | 2 (2) | 1 (1)
MEDICAL EXAM (Investigations) | 23 (33) | 22 (34)
MEDICATION ADJUSTMENT (Cardiac disorders) | 1 (1) | 0 (0)
MEGACOLON (Gastrointestinal disorders) | 1 (1) | 0 (0)
MENINGITIS (Nervous system disorders) | 1 (1) | 0 (0)
MESENTERIC ISCHEMIA (Gastrointestinal disorders) | 2 (2) | 0 (0)
METABOLIC ACIDOSIS (Renal and urinary disorders) | 1 (1) | 0 (0)
MITRAL REGURGITATION (Cardiac disorders) | 0 (0) | 1 (2)
MITRAL VALVE REPLACEMENT (Cardiac disorders) | 1 (1) | 0 (0)
MOTOR VEHICLE ACCIDENT (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
MRSA INFECTION (Infections and infestations) | 3 (3) | 1 (1)
MULTIPLE INFIRMITIES OF AGING (General disorders) | 0 (0) | 1 (1)
MULTIPLE ORGAN FAILURE (General disorders) | 3 (4) | 3 (3)
MYASTHENIA GRAVIS (Nervous system disorders) | 0 (0) | 1 (1)
MYELOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 67 (79) | 66 (83)
MYOCARDIAL INFARCTION (Nervous system disorders) | 1 (1) | 0 (0)
MYOCARDIAL INFECTION (Cardiac disorders) | 1 (1) | 1 (1)
MYOCLONIA (Nervous system disorders) | 0 (0) | 1 (1)
MYOMA (Reproductive system and breast disorders) | 1 (1) | 0 (0)
MYOPATHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 5 (5) | 1 (1)
NECK CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
NEPHRECTOMY (Surgical and medical procedures) | 0 (0) | 1 (1)
NEURONITIS (Nervous system disorders) | 0 (0) | 1 (1)
NEUROPATHY (Endocrine disorders) | 0 (0) | 1 (2)
NEUROPATHY (Nervous system disorders) | 3 (3) | 0 (0)
NON-CALCULOUS CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
OBSTRUCTIVE UROPATHY (Renal and urinary disorders) | 0 (0) | 1 (1)
OBTURATIVE SUPPURATIVE GANGRENOUSE CALCULOUS CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
OEDEMA (Cardiac disorders) | 1 (1) | 0 (0)
OPISTHORCHOSIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
OPISTHORCHOSIS (Infections and infestations) | 0 (0) | 1 (1)
OPTIC ATROPHY (Eye disorders) | 0 (0) | 1 (2)
ORTHOPNEA (Cardiac disorders) | 0 (0) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 7 (7) | 10 (12)
OSTEOCHONDROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
OSTEOMYELITIS (Infections and infestations) | 0 (0) | 1 (1)
OSTEOMYELITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
OVERACTIVE BLADDER (Renal and urinary disorders) | 1 (1) | 0 (0)
PACEMAKER IMPLANT (Cardiac disorders) | 0 (0) | 1 (1)
PALPITATIONS (Cardiac disorders) | 2 (2) | 1 (1)
PANCREATIC CANCER (Endocrine disorders) | 1 (1) | 0 (0)
PANCREATIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
PANCREATIC MASS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PANCREATITIS (Endocrine disorders) | 3 (3) | 2 (3)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 2 (2)
PANCREATITIS (Hepatobiliary disorders) | 1 (1) | 7 (9)
PANCYTOPENIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
PARASTHESIA (Nervous system disorders) | 2 (2) | 1 (1)
PARKINSON'S DISEASE (Nervous system disorders) | 1 (1) | 0 (0)
PAROTID GLAND CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PATHOLOGY OF ENDOMETRIUM (Reproductive system and breast disorders) | 1 (1) | 0 (0)
PENILE BLEEDING (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PERCUTANEOUS CORONARY INTERVENTION (Cardiac disorders) | 1 (1) | 0 (0)
PERICARDITIS (Cardiac disorders) | 0 (0) | 2 (2)
PERIPHERAL ARTERIAL DISEASE (Vascular disorders) | 6 (11) | 1 (1)
PERIPHERAL VASCULAR DISEASE (Vascular disorders) | 0 (0) | 1 (1)
PERITONITIS (Gastrointestinal disorders) | 2 (2) | 1 (1)
PERITONITIS (Infections and infestations) | 0 (0) | 1 (1)
PHLEBOTHROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 9 (12)
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 2 (2)
PNEUMONIA (Renal and urinary disorders) | 1 (1) | 0 (0)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 75 (83) | 76 (87)
POLYMYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
POLYP REMOVAL (Gastrointestinal disorders) | 1 (1) | 0 (0)
POLYPS (Gastrointestinal disorders) | 2 (2) | 0 (0)
POLYPS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 0 (0)
POLYPS (Reproductive system and breast disorders) | 1 (1) | 0 (0)
POST-MENOPAUSAL BLEEDING (Reproductive system and breast disorders) | 1 (1) | 0 (0)
PRE-CANCEROUS TUMOR SURGERY, LEFT TEMPORAL LEVEL. (Surgical and medical procedures) | 0 (0) | 1 (1)
PREVENTIVE TREATMENT (Surgical and medical procedures) | 1 (1) | 0 (0)
PROCTITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
PROPHYLACTIC THERAPY (Cardiac disorders) | 1 (1) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
PROSTATE CANCER (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PROSTATE SURGERY (Surgical and medical procedures) | 2 (2) | 1 (1)
PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 5 (5) | 2 (2)
PROSTATITIS (Renal and urinary disorders) | 0 (0) | 1 (1)
PROSTATITIS (Reproductive system and breast disorders) | 1 (1) | 0 (0)
PSYCHOSIS (Psychiatric disorders) | 1 (1) | 0 (0)
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY EDEMA (Cardiac disorders) | 3 (4) | 3 (5)
PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 8 (12) | 10 (11)
PULMONARY EMBOLISM (Cardiac disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 8 (8)
PULMONARY EMBOLUS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PULMONARY OVERLOAD (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 1 (1)
PURPURA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
PYELOCYSTITIS (Renal and urinary disorders) | 0 (0) | 2 (2)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 1 (1)
PYELONEPHRITIS (Renal and urinary disorders) | 1 (1) | 2 (2)
RADIATION (Surgical and medical procedures) | 0 (0) | 1 (1)
RADIOFREQUENCY ABLATION (Cardiac disorders) | 1 (1) | 1 (1)
RADIOFREQUENCY ABLATION (Surgical and medical procedures) | 0 (0) | 2 (2)
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
RECTAL PROLAPSE SURGERY (Gastrointestinal disorders) | 0 (0) | 1 (1)
RECTOVESICAL FISTULA (Gastrointestinal disorders) | 1 (1) | 0 (0)
RECTUS HEMATOMA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
REMOVAL OF ADHESIONS (Gastrointestinal disorders) | 1 (1) | 0 (0)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 1 (1) | 1 (1)
RENAL MASS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
RESECTION OF CUBITAL (Surgical and medical procedures) | 1 (1) | 0 (0)
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
RESPIRATORY FAILURE (Cardiac disorders) | 1 (1) | 2 (2)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 10 (10)
RESPIRATORY INSUFFICIENCY (Renal and urinary disorders) | 1 (1) | 0 (0)
RESPIRATORY INSUFFICIENCY (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
RESPIRATORY TRACT INFECTION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
RETINAL ANGIOPATHY (Eye disorders) | 0 (0) | 1 (1)
RETINAL DETACHMENT (Eye disorders) | 0 (0) | 1 (1)
RETINOPATHY (Eye disorders) | 0 (0) | 1 (1)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
RUPTURED ESOPHAGUS (Gastrointestinal disorders) | 0 (0) | 1 (1)
SALMONELLOSIS (Infections and infestations) | 1 (1) | 0 (0)
SCIATICA (Nervous system disorders) | 1 (1) | 0 (0)
SCLERODERMA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SCLERODERMA (Renal and urinary disorders) | 0 (0) | 1 (1)
SCLERODERMA (Vascular disorders) | 1 (2) | 0 (0)
SCLEROTIC METASTASIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SECONDARY TO ANTIARRHYTHMIC MEDICATION (Cardiac disorders) | 0 (0) | 1 (1)
SEIZURE (Nervous system disorders) | 4 (5) | 1 (1)
SEPSIS (General disorders) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 15 (15) | 16 (16)
SEPSIS (Renal and urinary disorders) | 1 (1) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 5 (5) | 3 (3)
SEPTIC SHOCK (Nervous system disorders) | 1 (1) | 0 (0)
SHINGLES (Endocrine disorders) | 1 (1) | 0 (0)
SHORTNESS OF BREATH (Cardiac disorders) | 1 (1) | 2 (2)
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 17 (19) | 22 (26)
SHOT (Cardiac disorders) | 0 (0) | 1 (1)
SHOULDER INJURY (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
SHOULDER SURGERY (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
SICCA SYNDROME (Immune system disorders) | 1 (1) | 0 (0)
SICK SINUS SYNDROME (Cardiac disorders) | 1 (2) | 2 (2)
SINUS CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SINUS NODE DISEASE (Cardiac disorders) | 0 (0) | 1 (1)
SINUSITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SKIN CANCER (Infections and infestations) | 1 (1) | 0 (0)
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 5 (5)
SKIN DISEASE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SKIN LACERATION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SKIN LESION (Infections and infestations) | 0 (0) | 1 (1)
SKULL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SMALL BOWEL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
SPINAL STENOSIS (Nervous system disorders) | 2 (2) | 1 (1)
SPINAL STENOSIS (Surgical and medical procedures) | 1 (1) | 1 (1)
SPINAL SURGERY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
STENT GRAFT (Cardiac disorders) | 0 (0) | 1 (1)
STENT RESTENOSIS (Surgical and medical procedures) | 1 (1) | 0 (0)
STERNUM DIASTASIS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
STOMACH CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
STROKE (Cardiac disorders) | 2 (2) | 3 (3)
STROKE (Nervous system disorders) | 57 (65) | 71 (80)
STROKE (Surgical and medical procedures) | 1 (1) | 0 (0)
SUBUNGUAL AND THECAL WHITLOW PANARICIUM OF THE LEFT HAND (Infections and infestations) | 1 (1) | 0 (0)
SUPRATHERAPEUTIC INR (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
SURGICAL PROCEDURE (Cardiac disorders) | 1 (1) | 0 (0)
SYNCOPE (Cardiac disorders) | 1 (1) | 1 (1)
SYNCOPE (Endocrine disorders) | 1 (1) | 0 (0)
SYNCOPE (General disorders) | 1 (1) | 0 (0)
SYNCOPE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 28 (30) | 21 (24)
TACHYCARDIA (Cardiac disorders) | 7 (7) | 5 (5)
TEE (Surgical and medical procedures) | 1 (1) | 0 (0)
THROAT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
THROMBOEMBOLISM (Cardiac disorders) | 1 (1) | 0 (0)
THROMBOEMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (1)
THROMBOEMBOLISM (Vascular disorders) | 1 (1) | 1 (1)
THROMBOSIS (Vascular disorders) | 2 (3) | 1 (3)
THYROIDECTOMY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
TOE AMPUTATION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
TOE AMPUTATION (Surgical and medical procedures) | 0 (0) | 1 (1)
TOOTH ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
TOOTHACHE (Infections and infestations) | 0 (0) | 1 (1)
TOXIC ALLERGIC ALVEOLITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
TOXIC PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
TRANSIENT ISCHEMIC ATTACK (Cardiac disorders) | 1 (2) | 2 (2)
TRANSIENT ISCHEMIC ATTACK (Nervous system disorders) | 7 (8) | 8 (9)
TRANSURETHRAL PROSTATIC RESECTION (Surgical and medical procedures) | 1 (1) | 0 (0)
TRAUMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
TREMOR (Nervous system disorders) | 1 (1) | 3 (3)
TRICUSPID REGURGITATION (Cardiac disorders) | 0 (0) | 1 (1)
TUMOR REMOVAL (Surgical and medical procedures) | 1 (1) | 1 (1)
ULCER (Gastrointestinal disorders) | 2 (2) | 1 (1)
ULCER (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
ULCER (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
ULCER (Vascular disorders) | 0 (0) | 1 (1)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 1 (1) | 1 (2)
UPPER RESPIRATORY INFECTION (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
URETER STONE (Renal and urinary disorders) | 1 (1) | 0 (0)
URETHRITIS (Renal and urinary disorders) | 0 (0) | 1 (1)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 3 (3) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Renal and urinary disorders) | 16 (22) | 18 (18)
URINARY TRACT STONES (Renal and urinary disorders) | 1 (1) | 2 (2)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
UTERINE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
UTERINE PROLAPSE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
UTERINE TUMOR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
VAGINITIS (Reproductive system and breast disorders) | 1 (1) | 0 (0)
VALVE REPLACEMENT (Cardiac disorders) | 1 (1) | 0 (0)
VALVE REPLACEMENT (Surgical and medical procedures) | 0 (0) | 2 (2)
VARICOSE VEINS (Vascular disorders) | 1 (1) | 0 (0)
VENOUS INSUFFICIENCY (Vascular disorders) | 0 (0) | 2 (2)
VENOUS STASIS (Vascular disorders) | 1 (1) | 0 (0)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 0 (0) | 3 (3)
VERTEBROBASILAR INSUFFICIENCY (Nervous system disorders) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 2 (2) | 1 (1)
VERTIGO (Nervous system disorders) | 1 (1) | 1 (1)
VISION CHANGES (Eye disorders) | 0 (0) | 1 (1)
VOLUME OVERLOAD (Vascular disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 2 (2) | 2 (2)
WARFARIN ALLERGIC REACTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
WARFARIN OVERDOSE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
WEAKNESS (Gastrointestinal disorders) | 0 (0) | 1 (1)
WEAKNESS (General disorders) | 2 (2) | 7 (7)
WEAKNESS (Nervous system disorders) | 3 (3) | 1 (1)
WEIGHT GAIN (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
WORSENING HF (Cardiac disorders) | 1 (1) | 1 (2)
WOUND INFECTION (Infections and infestations) | 2 (2) | 3 (3)
XERODERMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=1723) | Spironolactone (N=1722)
ABDOMINAL PAIN (Cardiac disorders) | 0 (0) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 28 (31) | 31 (34)
ABDOMINAL PAIN (Hepatobiliary disorders) | 1 (1) | 2 (2)
ABDOMINAL PAIN (Musculoskeletal and connective tissue disorders) | 3 (4) | 6 (6)
ABNORMAL BMP (General disorders) | 5 (9) | 1 (1)
ABNORMAL VAGINAL BLEEDING (Reproductive system and breast disorders) | 2 (2) | 3 (3)
ABSCESS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
ACUTE RESPIRATORY DISEASE (Respiratory, thoracic and mediastinal disorders) | 15 (17) | 9 (9)
ALLERGY (Immune system disorders) | 11 (12) | 11 (12)
ALTERED MENTAL STATUS (Nervous system disorders) | 9 (9) | 12 (12)
ANEMIA (Blood and lymphatic system disorders) | 44 (48) | 41 (45)
ANEMIA (Cardiac disorders) | 2 (2) | 0 (0)
ANEURYSM (Cardiac disorders) | 3 (3) | 0 (0)
ANGINA (Cardiac disorders) | 2 (2) | 0 (0)
ANGIOGRAPHY (Surgical and medical procedures) | 2 (2) | 0 (0)
ANGIOPATHY (Vascular disorders) | 2 (2) | 0 (0)
ANKLE INJURY (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
ANXIETY (Nervous system disorders) | 3 (3) | 1 (1)
ANXIETY (Psychiatric disorders) | 3 (3) | 4 (4)
ARM INJURY (General disorders) | 2 (2) | 0 (0)
ARM INJURY (Musculoskeletal and connective tissue disorders) | 14 (15) | 10 (10)
ARRHYTHMIA (Cardiac disorders) | 16 (18) | 10 (13)
ARTERIAL STENOSIS (Cardiac disorders) | 2 (2) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 (5) | 8 (14)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 11 (12) | 10 (10)
ASTHENIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 9 (9)
ATAXIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
ATAXIA (Nervous system disorders) | 2 (2) | 5 (5)
ATHEROSCLEROSIS (Cardiac disorders) | 2 (2) | 3 (4)
ATHEROSCLEROSIS (Nervous system disorders) | 1 (1) | 2 (2)
ATHEROSCLEROSIS (Vascular disorders) | 0 (0) | 4 (4)
ATRIAL FIBRILLATION (Cardiac disorders) | 85 (123) | 74 (97)
ATRIAL FLUTTER (Cardiac disorders) | 5 (6) | 7 (9)
AV BLOCK (Cardiac disorders) | 0 (0) | 2 (2)
BACK INJURY (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 64 (74) | 67 (76)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
BLADDER TUMOR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
BLEEDING (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
BLEEDING IN EYE (Eye disorders) | 1 (1) | 7 (8)
BLOOD IN STOOL (Gastrointestinal disorders) | 3 (3) | 0 (0)
BLURRED VISION (Eye disorders) | 9 (9) | 5 (5)
BODY ACHES (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
BODY PAIN (Musculoskeletal and connective tissue disorders) | 9 (11) | 9 (9)
BRADYCARDIA (Cardiac disorders) | 8 (8) | 20 (22)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
BREAST PAIN (Reproductive system and breast disorders) | 5 (5) | 18 (18)
BREAST TENDERNESS (Reproductive system and breast disorders) | 0 (0) | 2 (2)
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 64 (69) | 63 (75)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 2 (2)
BRUISE (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
BRUISE (Musculoskeletal and connective tissue disorders) | 5 (7) | 1 (1)
BRUISE (Skin and subcutaneous tissue disorders) | 9 (9) | 11 (12)
BUNDLE BRANCH BLOCK (Cardiac disorders) | 0 (0) | 2 (2)
BURSITIS (Musculoskeletal and connective tissue disorders) | 8 (8) | 2 (2)
BUTTOCK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
C-DIFF INFECTION (Infections and infestations) | 5 (5) | 0 (0)
CANCER REMOVAL (Surgical and medical procedures) | 0 (0) | 2 (2)
CARDIOVERSION (Cardiac disorders) | 4 (5) | 2 (2)
CARPEL TUNNEL RELEASE (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
CARPEL TUNNEL SYNDROME (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
CARPEL TUNNEL SYNDROME (Nervous system disorders) | 3 (5) | 1 (1)
CATARACTS (Eye disorders) | 17 (21) | 18 (21)
CELLULITIS (Infections and infestations) | 11 (11) | 2 (2)
CELLULITIS (Skin and subcutaneous tissue disorders) | 20 (20) | 18 (22)
CHEMOTHERAPY (Surgical and medical procedures) | 2 (3) | 0 (0)
CHEST CONGESTION (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
CHEST PAIN (Cardiac disorders) | 102 (130) | 80 (102)
CHEST PAIN (Musculoskeletal and connective tissue disorders) | 8 (8) | 11 (12)
CHILLS (General disorders) | 0 (0) | 2 (3)
CHOLECYSTITIS (Hepatobiliary disorders) | 4 (4) | 5 (5)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 14 (15) | 10 (12)
CLAUDICATION (Vascular disorders) | 2 (2) | 1 (1)
COLD EXTREMITIES (Vascular disorders) | 4 (4) | 1 (1)
COLD SYMPTOMS (General disorders) | 3 (3) | 0 (0)
COLITIS (Gastrointestinal disorders) | 3 (3) | 4 (4)
COLONOSCOPY (Surgical and medical procedures) | 2 (2) | 0 (0)
CONCUSSION (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
CONFUSION (Nervous system disorders) | 9 (10) | 5 (5)
CONJUCTIVITIS (Eye disorders) | 5 (5) | 8 (8)
CONSTIPATION (Gastrointestinal disorders) | 25 (26) | 28 (31)
CORONARY ARTERY DISEASE (Cardiac disorders) | 3 (3) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 44 (53) | 44 (47)
CYST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (14) | 18 (19)
CYST (Renal and urinary disorders) | 2 (2) | 0 (0)
CYSTOSCOPY (Renal and urinary disorders) | 2 (2) | 0 (0)
DECREASED APPETITE (Gastrointestinal disorders) | 8 (8) | 10 (10)
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 4 (4) | 2 (2)
DEHYDRATION (Gastrointestinal disorders) | 2 (2) | 0 (0)
DEHYDRATION (General disorders) | 4 (4) | 13 (13)
DEMENTIA (Nervous system disorders) | 2 (2) | 2 (2)
DENTAL ABSCESS (Infections and infestations) | 2 (2) | 1 (1)
DEPRESSION (Psychiatric disorders) | 16 (16) | 20 (20)
DERMATITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
DERMATITIS (Skin and subcutaneous tissue disorders) | 27 (29) | 25 (26)
DESTABILIZATION OF BLOOD PRESSURE (Cardiac disorders) | 2 (2) | 0 (0)
DEVICE CHANGE (Cardiac disorders) | 3 (3) | 4 (4)
DIABETES (Endocrine disorders) | 37 (40) | 38 (42)
DIABETES (Renal and urinary disorders) | 0 (0) | 2 (2)
DIAPHORESIS (General disorders) | 2 (2) | 0 (0)
DIARRHEA (Gastrointestinal disorders) | 74 (83) | 79 (88)
DIVERTICULITIS (Gastrointestinal disorders) | 3 (3) | 2 (2)
DIZZINESS (Cardiac disorders) | 3 (3) | 2 (2)
DIZZINESS (General disorders) | 35 (44) | 34 (35)
DIZZINESS (Nervous system disorders) | 54 (70) | 64 (75)
DORSOPATHY (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
DROWSINESS (Nervous system disorders) | 2 (2) | 3 (3)
DRY EYES (Eye disorders) | 1 (1) | 2 (2)
DUODENITIS (Gastrointestinal disorders) | 1 (1) | 2 (2)
DYSLIPIDEMIA (Cardiac disorders) | 2 (2) | 1 (1)
DYSLIPIDEMIA (General disorders) | 16 (18) | 13 (13)
DYSLIPIDEMIA (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 4 (5) | 2 (2)
DYSPHAGIA (Gastrointestinal disorders) | 4 (4) | 4 (4)
DYSPNEA (Cardiac disorders) | 37 (44) | 31 (32)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
DYSURIA (Renal and urinary disorders) | 7 (7) | 6 (6)
EAR ACHE (Ear and labyrinth disorders) | 2 (2) | 2 (2)
EAR INFECTION (Ear and labyrinth disorders) | 7 (7) | 6 (6)
EAR INFECTION (Infections and infestations) | 3 (3) | 1 (1)
EAR PAIN (Ear and labyrinth disorders) | 0 (0) | 3 (3)
EDEMA (Cardiac disorders) | 3 (3) | 4 (4)
EDEMA (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
ELEVATED BILIRUBIN (Hepatobiliary disorders) | 0 (0) | 2 (2)
ELEVATED BNP (Cardiac disorders) | 2 (2) | 0 (0)
ELEVATED BUN (Renal and urinary disorders) | 3 (3) | 4 (4)
ELEVATED CARDIAC ENZYMES (Cardiac disorders) | 5 (5) | 9 (9)
ELEVATED CREATININE (Renal and urinary disorders) | 47 (50) | 60 (77)
ELEVATED INR (Blood and lymphatic system disorders) | 2 (3) | 4 (4)
ELEVATED LIVER ENZYMES (Hepatobiliary disorders) | 4 (4) | 5 (6)
ELEVATED LIVER ENZYMES (Renal and urinary disorders) | 2 (2) | 1 (2)
ELEVATED PSA (Reproductive system and breast disorders) | 0 (0) | 2 (2)
EMOTIONAL LABILITY (Psychiatric disorders) | 2 (2) | 4 (4)
ENCEPHALOPATHY (Nervous system disorders) | 8 (8) | 6 (6)
EPIGASTRIC PAIN (Gastrointestinal disorders) | 3 (3) | 1 (1)
EPISTAXIS (Vascular disorders) | 21 (21) | 19 (27)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 4 (4) | 3 (3)
ERYTHROCYTOSIS (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
ESOPHAGITIS (Gastrointestinal disorders) | 3 (3) | 0 (0)
EXTRASYSTOLE (Cardiac disorders) | 7 (7) | 7 (8)
EYE PAIN (Eye disorders) | 2 (3) | 3 (4)
EYELID CYSTS (Eye disorders) | 0 (0) | 2 (2)
FALL (Injury, poisoning and procedural complications) | 4 (5) | 3 (3)
FALL (Musculoskeletal and connective tissue disorders) | 12 (12) | 15 (17)
FALL (Nervous system disorders) | 4 (7) | 2 (3)
FATIGUE (Cardiac disorders) | 2 (2) | 1 (1)
FATIGUE (General disorders) | 17 (18) | 7 (7)
FATTY HEPATOSIS (Hepatobiliary disorders) | 2 (2) | 1 (1)
FEVER (General disorders) | 8 (8) | 3 (3)
FEVER (Infections and infestations) | 2 (2) | 5 (5)
FLATULENCE (Gastrointestinal disorders) | 2 (2) | 2 (2)
FLU LIKE SYMPTOMS (General disorders) | 2 (2) | 1 (1)
FLUID RETENTION (General disorders) | 0 (0) | 2 (2)
FOOT INJURY (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
FOOT PAIN (Musculoskeletal and connective tissue disorders) | 6 (8) | 7 (7)
FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
FRACTURE (Musculoskeletal and connective tissue disorders) | 33 (34) | 28 (30)
GALLSTONES (Hepatobiliary disorders) | 5 (5) | 7 (10)
GASTRIC REFLUX (Gastrointestinal disorders) | 7 (7) | 3 (3)
GASTRITIS (Gastrointestinal disorders) | 58 (59) | 52 (59)
GASTROENTERITIS (Gastrointestinal disorders) | 14 (14) | 6 (6)
GI BLEED (Gastrointestinal disorders) | 8 (8) | 11 (11)
GI DISTRESS (Gastrointestinal disorders) | 6 (6) | 7 (7)
GLAUCOMA (Eye disorders) | 2 (2) | 3 (3)
GOITER (Endocrine disorders) | 2 (2) | 7 (7)
GONITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
GOUT (Musculoskeletal and connective tissue disorders) | 36 (48) | 34 (38)
GYNECOMASTIA (Endocrine disorders) | 0 (0) | 6 (6)
GYNECOMASTIA (Reproductive system and breast disorders) | 7 (8) | 44 (45)
HAIR LOSS (Immune system disorders) | 1 (1) | 3 (3)
HAND INJURY (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
HAND PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4)
HAY FEVER (Immune system disorders) | 1 (1) | 2 (2)
HEAD INJURY (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
HEADACHE (Cardiac disorders) | 2 (2) | 2 (2)
HEADACHE (Nervous system disorders) | 90 (113) | 84 (98)
HEARING LOSS (Ear and labyrinth disorders) | 8 (9) | 4 (4)
HEART FAILURE (Cardiac disorders) | 135 (174) | 121 (150)
HEART VALVE CALCIFICATION (Cardiac disorders) | 3 (3) | 0 (0)
HEARTBURN (Cardiac disorders) | 1 (1) | 2 (2)
HEARTBURN (Gastrointestinal disorders) | 7 (7) | 7 (7)
HEMATEMESIS (Gastrointestinal disorders) | 1 (1) | 2 (2)
HEMATOMA (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
HEMATOMA (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (3)
HEMATURIA (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
HEMATURIA (Renal and urinary disorders) | 10 (10) | 11 (11)
HEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (6)
HEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 3 (3)
HEMORRHOIDS (Vascular disorders) | 0 (0) | 2 (2)
HERNIA (Musculoskeletal and connective tissue disorders) | 13 (14) | 6 (6)
HERNIA (Surgical and medical procedures) | 2 (2) | 0 (0)
HERPES SIMPLEX (Infections and infestations) | 1 (1) | 2 (2)
HIP PAIN (Musculoskeletal and connective tissue disorders) | 10 (10) | 17 (20)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
HOT FLASHES (Endocrine disorders) | 2 (2) | 1 (1)
HYPERCALCEMIA (General disorders) | 0 (0) | 2 (2)
HYPERCALCEMIA (Renal and urinary disorders) | 2 (2) | 0 (0)
HYPEREMIA (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
HYPERGLYCEMIA (Endocrine disorders) | 26 (29) | 21 (25)
HYPERKALEMIA (Cardiac disorders) | 0 (0) | 2 (2)
HYPERKALEMIA (Endocrine disorders) | 2 (2) | 1 (1)
HYPERKALEMIA (Metabolism and nutrition disorders) | 3 (4) | 5 (6)
HYPERKALEMIA (Renal and urinary disorders) | 96 (109) | 226 (273)
HYPERTENSIC CRISIS (Cardiac disorders) | 4 (4) | 0 (0)
HYPERTENSION (Cardiac disorders) | 145 (265) | 113 (219)
HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
HYPERTHERMIA (Infections and infestations) | 0 (0) | 2 (2)
HYPERTHYROIDISM (Endocrine disorders) | 2 (2) | 3 (3)
HYPERURICEMIA (Renal and urinary disorders) | 1 (1) | 4 (5)
HYPERVOLEMIA (Cardiac disorders) | 6 (9) | 7 (14)
HYPOGLYCEMIA (Endocrine disorders) | 19 (27) | 9 (9)
HYPOKALEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
HYPOKALEMIA (Renal and urinary disorders) | 29 (38) | 13 (17)
HYPONATREMIA (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
HYPONATREMIA (Renal and urinary disorders) | 0 (0) | 10 (12)
HYPOTENSION (Cardiac disorders) | 52 (59) | 71 (90)
HYPOTHYROIDISM (Endocrine disorders) | 8 (8) | 15 (15)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
INCREASED OF TSH (Endocrine disorders) | 2 (2) | 1 (1)
INFECTION (Infections and infestations) | 5 (5) | 8 (8)
INFLUENZA (General disorders) | 6 (6) | 2 (2)
INFLUENZA (Infections and infestations) | 71 (82) | 70 (80)
INFLUENZA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
INGROWN TOENAIL (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
INSOMNIA (Nervous system disorders) | 39 (55) | 29 (46)
IRON DEFICIENCY (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
IRON OVERLOAD (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
KIDNEY DISEASE (Renal and urinary disorders) | 68 (76) | 135 (182)
KIDNEY STONE (Renal and urinary disorders) | 8 (10) | 5 (6)
KNEE INJURY (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
KNEE PAIN (Musculoskeletal and connective tissue disorders) | 12 (12) | 20 (22)
LABYRINTHITIS (Ear and labyrinth disorders) | 0 (0) | 3 (3)
LACTOSE INTOLERANCE (Gastrointestinal disorders) | 2 (2) | 0 (0)
LEG CLAUDICATION (Vascular disorders) | 2 (2) | 1 (1)
LEG EDEMA (Cardiac disorders) | 3 (3) | 0 (0)
LEG INJURY (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
LEG PAIN (Musculoskeletal and connective tissue disorders) | 30 (31) | 29 (30)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 5 (5) | 2 (2)
LIMB EDEMA (Cardiac disorders) | 2 (2) | 2 (2)
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (3)
LOW HEMOGLOBIN (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
LOWER EXTREMITY EDEMA (Cardiac disorders) | 40 (44) | 36 (41)
LOWER EXTREMITY EDEMA (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
LOWER EXTREMITY EDEMA (Vascular disorders) | 3 (3) | 3 (3)
LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
LUNG MASS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
MACULAR DEGENERATION (Eye disorders) | 2 (2) | 2 (2)
MEMORY LOSS (Nervous system disorders) | 2 (2) | 7 (9)
MOUTH PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
MUSCLE INJURY (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
MUSCLE PAIN (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (6)
MUSCLE SPASM (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (2) | 2 (2)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
NAUSEA (Gastrointestinal disorders) | 34 (37) | 54 (57)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 5 (5) | 7 (7)
NEURALGIA (Nervous system disorders) | 1 (1) | 2 (2)
NEUROPATHY (Nervous system disorders) | 7 (7) | 4 (4)
NEUROSIS (Psychiatric disorders) | 13 (21) | 6 (8)
NOCTURIA (Renal and urinary disorders) | 2 (2) | 0 (0)
OLIGURIA (Renal and urinary disorders) | 2 (2) | 0 (0)
ONYCHOMYCOSIS (Infections and infestations) | 1 (1) | 2 (2)
ORTHOPNEA (Cardiac disorders) | 2 (2) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 14 (14) | 26 (27)
OSTEOCHONDROSIS (Musculoskeletal and connective tissue disorders) | 10 (10) | 14 (15)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
OTITIS (Ear and labyrinth disorders) | 0 (0) | 2 (2)
PALPITATIONS (Cardiac disorders) | 26 (29) | 25 (26)
PARAGEUSIA (Gastrointestinal disorders) | 2 (3) | 2 (2)
PARASTHESIA (Nervous system disorders) | 20 (24) | 23 (26)
PARKINSON'S DISEASE (Nervous system disorders) | 1 (1) | 2 (2)
PERICARDITIS (Cardiac disorders) | 1 (1) | 2 (2)
PERIPHERAL ARTERIAL DISEASE (Vascular disorders) | 0 (0) | 3 (3)
PERIPHERAL EDEMA (Cardiac disorders) | 4 (4) | 1 (1)
PHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (7)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 31 (32) | 44 (49)
POLYPS (Gastrointestinal disorders) | 2 (2) | 2 (2)
POLYPS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 9 (9)
POLYURIA (Renal and urinary disorders) | 4 (4) | 4 (4)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (4)
PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 6 (6) | 6 (6)
PROTEINURIA (Renal and urinary disorders) | 2 (2) | 4 (4)
PRURITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
PRURITIS (Skin and subcutaneous tissue disorders) | 8 (9) | 14 (14)
PSORIASIS (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (5)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
PULMONARY OVERLOAD (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4)
PURITIS (Skin and subcutaneous tissue disorders) | 3 (5) | 1 (1)
PYELONEPHRITIS (Renal and urinary disorders) | 8 (8) | 9 (9)
RADICULITIS (Nervous system disorders) | 7 (8) | 8 (8)
RASH (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 2 (2) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
RESPIRATORY TRACT INFECTION (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5)
RESTLESS LEG SYNDROME (Nervous system disorders) | 2 (2) | 1 (1)
RETINOPATHY (Eye disorders) | 0 (0) | 2 (2)
RHINITIS (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 10 (12)
RIB PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
SCIATICA (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
SCIATICA (Nervous system disorders) | 1 (1) | 7 (7)
SEASONAL ALLERGIES (Immune system disorders) | 0 (0) | 2 (2)
SEIZURE (Nervous system disorders) | 4 (4) | 3 (3)
SEPSIS (Infections and infestations) | 3 (3) | 0 (0)
SEXUALLY TRANSMITTED DISEASE (Infections and infestations) | 2 (2) | 0 (0)
SHINGLES (Infections and infestations) | 7 (7) | 10 (10)
SHORTNESS OF BREATH (Cardiac disorders) | 2 (4) | 3 (4)
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 34 (40) | 27 (30)
SHOULDER INJURY (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
SHOULDER INJURY (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 14 (14) | 9 (10)
SICK SINUS SYNDROME (Cardiac disorders) | 1 (1) | 4 (4)
SINUSITIS (Infections and infestations) | 4 (4) | 3 (3)
SINUSITIS (Respiratory, thoracic and mediastinal disorders) | 19 (21) | 14 (17)
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17 (22) | 14 (15)
SKIN LACERATION (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
SKIN LACERATION (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
SKIN LACERATION (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (6)
SKIN LESION (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
SKIN WOUND (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
SLEEP APNEA (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 9 (9)
SLEEP DISTURBANCE (Nervous system disorders) | 1 (1) | 2 (2)
SORE THROAT (Gastrointestinal disorders) | 0 (0) | 2 (2)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
STENOSING TENOSYNOVITIS (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
STOMACH ULCER (Gastrointestinal disorders) | 2 (2) | 1 (1)
STROKE (Nervous system disorders) | 10 (11) | 8 (11)
SUPRATHERAPEUTIC INR (Blood and lymphatic system disorders) | 3 (3) | 1 (2)
SWEATING (General disorders) | 2 (2) | 3 (3)
SYNCOPE (Nervous system disorders) | 24 (27) | 28 (28)
TACHYCARDIA (Cardiac disorders) | 20 (29) | 22 (25)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
THROMBOPHLEBITIS (Vascular disorders) | 6 (6) | 2 (2)
THRUSH (Infections and infestations) | 3 (3) | 1 (1)
THYROID NODULE (Endocrine disorders) | 2 (2) | 1 (1)
THYROID NODULE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
TINNITUS (Ear and labyrinth disorders) | 2 (2) | 5 (5)
TMJ DISORDER (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
TONGUE LESION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
TONSILLITIS (Infections and infestations) | 0 (0) | 2 (2)
TOOTH ABSCESS (Infections and infestations) | 2 (2) | 2 (2)
TOOTH EXTRACTION (Surgical and medical procedures) | 0 (0) | 3 (3)
TOOTHACHE (Musculoskeletal and connective tissue disorders) | 12 (13) | 8 (9)
TRANSIENT ISCHEMIC ATTACK (Nervous system disorders) | 11 (14) | 3 (3)
TREMOR (Nervous system disorders) | 5 (5) | 5 (5)
ULCER (Gastrointestinal disorders) | 4 (4) | 8 (8)
ULCER (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
ULCER (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3)
ULCER (Skin and subcutaneous tissue disorders) | 6 (7) | 4 (4)
ULCER (Vascular disorders) | 3 (4) | 2 (3)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 7 (7) | 4 (6)
UPPER RESPIRATORY INFECTION (Respiratory, thoracic and mediastinal disorders) | 78 (90) | 86 (98)
URETHRITIS (Gastrointestinal disorders) | 0 (0) | 2 (2)
URETHRITIS (Renal and urinary disorders) | 0 (0) | 2 (2)
URINARY HESITANCY (Renal and urinary disorders) | 2 (2) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 5 (6) | 7 (7)
URINARY RETENTION (Renal and urinary disorders) | 5 (5) | 10 (10)
URINARY TRACT INFECTION (Renal and urinary disorders) | 68 (84) | 60 (74)
URINARY TRACT STONES (Renal and urinary disorders) | 1 (1) | 2 (2)
URINARY URGENCY (Renal and urinary disorders) | 2 (2) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 2 (2) | 8 (9)
VARICOSE VEINS (Vascular disorders) | 5 (5) | 8 (10)
VENOUS INSUFFICIENCY (Vascular disorders) | 3 (4) | 10 (12)
VERTIGO (Ear and labyrinth disorders) | 16 (20) | 11 (11)
VERTIGO (Nervous system disorders) | 2 (2) | 1 (1)
VISION CHANGES (Eye disorders) | 2 (2) | 2 (2)
VISION LOSS (Eye disorders) | 3 (3) | 5 (5)
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
VOMITING (Gastrointestinal disorders) | 20 (20) | 20 (21)
WEAKNESS (Cardiac disorders) | 2 (2) | 0 (0)
WEAKNESS (Gastrointestinal disorders) | 2 (2) | 0 (0)
WEAKNESS (General disorders) | 35 (37) | 45 (53)
WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
WEAKNESS (Nervous system disorders) | 2 (2) | 2 (2)
WEIGHT GAIN (Metabolism and nutrition disorders) | 16 (17) | 15 (17)
WEIGHT LOSS (General disorders) | 1 (1) | 2 (2)
WEIGHT LOSS (Metabolism and nutrition disorders) | 8 (9) | 5 (7)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
WOUND INFECTION (Infections and infestations) | 2 (2) | 1 (1)
XEROSTOMIA (Gastrointestinal disorders) | 7 (7) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No